CLINICAL TRIAL: NCT03398148
Title: A Multicenter, Randomized, Double-Blind, Placebo Controlled Induction Study to Evaluate the Efficacy and Safety of Risankizumab in Subjects With Moderately to Severely Active Ulcerative Colitis
Brief Title: A Multicenter, Randomized, Double-Blind, Placebo Controlled Induction Study to Evaluate the Efficacy and Safety of Risankizumab in Participants With Moderately to Severely Active Ulcerative Colitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M16-067; 2016-004677-40 (EudraCT Number)
Record Dates: First submitted 2018-01-08; First posted 2018-01-12 (Actual); Results first posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Ulcerative Colitis (UC)
Keywords: ABBV-066; BI 655066
MeSH Terms: conditions — Colitis, Ulcerative | interventions — risankizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (15):
- Substudy 1, Induction Period 1: Double-blind Placebo IV (Placebo Comparator): Participants randomized to receive placebo for risankizumab administered by intravenous (IV) infusion.
  Interventions: Drug: placebo for risankizumab
- Substudy 1, Induction Period 1: Double-blind Risankizumab 600mg IV (Experimental): Participants randomized to receive risankizumab 600mg administered by intravenous (IV) infusion.
  Interventions: Drug: risankizumab IV
- Substudy 1, Induction Period 1: Double-blind Risankizumab 1200mg IV (Experimental): Participants randomized to receive risankizumab 1200mg administered by intravenous (IV) infusion.
  Interventions: Drug: risankizumab IV
- Substudy 1, Induction Period 1: Double-blind Risankizumab 1800mg IV (Experimental): Participants randomized to receive risankizumab 1800mg administered by intravenous (IV) infusion.
  Interventions: Drug: risankizumab IV
- Substudy 1, Induction Period 1: Open-label Risankizumab 1800mg IV (Experimental): Participants receive risankizumab 1800mg administered by intravenous (IV) infusion.
  Interventions: Drug: risankizumab IV
- Substudy 1, Induction Period 2: Double-blind Risankizumab 180mg SC (Experimental): Participants who received risankizumab with inadequate response in Induction 1 randomized to receive risankizumab 180mg administered by subcutaneous (SC) injection in Induction 2.
  Interventions: Drug: risankizumab SC
- Substudy 1, Induction Period 2: Double-blind Risankizumab 360mg SC (Experimental): Participants who received risankizumab with inadequate response in Induction 1 randomized to receive risankizumab 360mg administered by subcutaneous (SC) injection in Induction 2.
  Interventions: Drug: risankizumab SC
- Substudy 1, Induction Period 2: Double-blind Risankizumab 1800mg IV (Experimental): Participants who received risankizumab with inadequate response in Induction 1 randomized to receive risankizumab 1800mg administered by intravenous (IV) infusion in Induction 2.
  Interventions: Drug: risankizumab IV
- Substudy 1, Induction Period 2: Double-blind Risankizumab 1800mg IV Pbo (Experimental): Participants who received placebo with inadequate response in Induction 1 receive risankizumab 1800mg administered by intravenous (IV) infusion in Induction 2.
  Interventions: Drug: risankizumab IV
- Substudy 2, Induction Period 1: Double-blind Placebo IV (Placebo Comparator): Participants randomized to receive placebo for risankizumab administered by intravenous (IV) infusion.
  Interventions: Drug: placebo for risankizumab
- Substudy 2, Induction Period 1: Double-blind Risankizumab 1200mg IV (Experimental): Participants randomized to receive risankizumab 1200mg administered by intravenous (IV) infusion.
  Interventions: Drug: risankizumab IV
- Substudy 2, Induction Period 2: Double-blind Risankizumab 180mg SC (Experimental): Participants who received risankizumab with inadequate response in Induction 1 randomized to receive risankizumab 180mg administered by subcutaneous (SC) injection in Induction 2.
  Interventions: Drug: risankizumab SC
- Substudy 2, Induction Period 2: Double-blind Risankizumab 360mg SC (Experimental): Participants who received risankizumab with inadequate response in Induction 1 randomized to receive risankizumab 360mg administered by subcutaneous (SC) injection in Induction 2.
  Interventions: Drug: risankizumab SC
- Substudy 2, Induction Period 2: Double-blind Risankizumab 1200mg IV (Experimental): Participants who received risankizumab with inadequate response in Induction 1 randomized to receive risankizumab 1200mg administered by intravenous (IV) infusion in Induction 2.
  Interventions: Drug: risankizumab IV
- Substudy 2, Induction Period 2: Double-blind Risankizumab 1200mg IV Pbo (Experimental): Participants who received placebo with inadequate response in Induction 1 randomized to receive risankizumab 1200mg administered by intravenous (IV) infusion in Induction 2.
  Interventions: Drug: risankizumab IV

INTERVENTIONS:
Drug: risankizumab IV — risankizumab intravenous (IV) infusion
  Other Names: ABBV-066; BI 655066
  Arms: Substudy 1, Induction Period 1: Double-blind Risankizumab 1200mg IV; Substudy 1, Induction Period 1: Double-blind Risankizumab 1800mg IV; Substudy 1, Induction Period 1: Double-blind Risankizumab 600mg IV; Substudy 1, Induction Period 1: Open-label Risankizumab 1800mg IV; Substudy 1, Induction Period 2: Double-blind Risankizumab 1800mg IV; Substudy 1, Induction Period 2: Double-blind Risankizumab 1800mg IV Pbo; Substudy 2, Induction Period 1: Double-blind Risankizumab 1200mg IV; Substudy 2, Induction Period 2: Double-blind Risankizumab 1200mg IV; Substudy 2, Induction Period 2: Double-blind Risankizumab 1200mg IV Pbo
Drug: placebo for risankizumab — placebo for risankizumab
  Arms: Substudy 1, Induction Period 1: Double-blind Placebo IV; Substudy 2, Induction Period 1: Double-blind Placebo IV
Drug: risankizumab SC — risankizumab subcutaneous (SC) injection
  Other Names: ABBV-066; BI 655066
  Arms: Substudy 1, Induction Period 2: Double-blind Risankizumab 180mg SC; Substudy 1, Induction Period 2: Double-blind Risankizumab 360mg SC; Substudy 2, Induction Period 2: Double-blind Risankizumab 180mg SC; Substudy 2, Induction Period 2: Double-blind Risankizumab 360mg SC

SUMMARY:
The objectives of Sub-Study 1 are to evaluate the efficacy, safety, and pharmacokinetics of risankizumab as induction treatment in subjects with moderately to severely active ulcerative colitis (UC), and to identify the appropriate induction dose of risankizumab for further evaluation in Sub-Study 2.

The objective of Sub-Study 2 is to evaluate the efficacy and safety of risankizumab compared to placebo in inducing clinical remission in subjects with moderately to severely active UC.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged >=18 to <= 80 years at the Baseline Visit. Where locally permissible, subjects 16 to < 18 years of age who meet the definition of Tanner stage 5 for development at the Baseline Visit.
* Confirmed diagnosis of ulcerative colitis (UC) for at least 3 months prior to Baseline.
* Active UC as assessed by Adapted Mayo Score and Endoscopic Subscore.
* Demonstrated intolerance or inadequate response to conventional therapy and tofacitinib (not a biologic) and one or more biologic therapies.
* Females must be postmenopausal for more than 1 year or surgically sterile or practicing specific forms of birth control.

Exclusion Criteria:

* Participant with a current diagnosis of Crohn's disease (CD), inflammatory bowel disease-unclassified (IBD-U) or a history of radiation colitis or ischemic colitis.
* Participant receiving prohibited medications and treatment.
* Extent of inflammatory disease limited to the rectum as assessed by screening endoscopy.
* Participant with currently known complications of UC (e.g., megacolon).
* No known active Coronavirus Disease - 2019 (COVID-19) infection.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1558 (Actual)
Dates: Start 2018-03-07 (Actual); Primary Completion 2022-11-09 (Actual); Study Completion 2023-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (430):
- United States (82):
  - Southern California Res. Ctr. /ID# 169660, Coronado, California
  - Hoag Memorial Hosp Presbyterian /ID# 218348, Irvine, California
  - UC San Diego Health System /ID# 160452, La Jolla, California
  - United Medical Doctors /ID# 158528, Los Alamitos, California
  - Gastrointestinal Biosciences Clinical Trials, LLC /ID# 200931, Los Angeles, California
  - UCSF Center for Colitis and Crohn's Disease /ID# 201210, San Francisco, California
  - Cedars-Sinai Medical Center-West Hollywood /ID# 163851, West Hollywood, California
  - Peak Gastroenterology Associates, PC /ID# 165841, Colorado Springs, Colorado
  - Rocky Mountain Pediatric Gastroenterology /ID# 207174, Lone Tree, Colorado
  - Medical Research Center of CT /ID# 160311, Hamden, Connecticut
  - Yale Univ Digestive Diseases /ID# 213179, New Haven, Connecticut
  - South Lake Pain Institute, Inc /ID# 162878, Clermont, Florida
  - Ctr for Advanced Gastroenterol /ID# 202811, Maitland, Florida
  - University of Miami /ID# 160471, Miami, Florida
  - Coral Research Clinic /ID# 158584, Miami, Florida
  - South Florida Research Ph I-IV, Inc. /ID# 161848, Miami, Florida
  - Gastroenterology Group Naples /ID# 165212, Naples, Florida
  - Advanced Research Institute, Inc /ID# 161938, New Port Richey, Florida
  - Advent Health /ID# 160433, Orlando, Florida
  - Endoscopic Research, Inc. /ID# 206711, Orlando, Florida
  - Omega Research Group /ID# 203059, Orlando, Florida
  - Lenus Research & Medical Group /ID# 169730, Sweetwater, Florida
  - Clinical Research Trials of Florida, Inc. /ID# 201783, Tampa, Florida
  - AdventHealth Tampa /ID# 170503, Tampa, Florida
  - Gastroenterology Associates of Central Georgia, LLC /ID# 160523, Macon, Georgia
  - Atlanta Gastroenterology Spec /ID# 161372, Suwanee, Georgia
  - The University of Chicago Medical Center /ID# 160521, Chicago, Illinois
  - DM Clinical Research/Southwest /ID# 165012, Oak Lawn, Illinois
  - Indiana University /ID# 167252, Indianapolis, Indiana
  - Univ Kansas Med Ctr /ID# 226602, Kansas City, Kansas
  - Cotton-O'Neil Clinical Res Ctr /ID# 160412, Topeka, Kansas
  - Robley Rex VA Medical Center /ID# 218648, Louisville, Kentucky
  - Houma Digestive Health Special /ID# 158317, Houma, Louisiana
  - Delricht Research /ID# 206815, New Orleans, Louisiana
  - Nola Research Works, LLC /ID# 161368, New Orleans, Louisiana
  - Louisana Research Center, LLC /ID# 201204, Shreveport, Louisiana
  - Massachusetts General Hospital - Crohn's and Colitis Center /ID# 164255, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center Michigan Medicine /ID# 158524, Ann Arbor, Michigan
  - Clin Res Inst of Michigan, LLC /ID# 160327, Chesterfield, Michigan
  - Mayo Clinic - Rochester /ID# 200458, Rochester, Minnesota
  - Quality Clinical Research Inc. /ID# 167313, Omaha, Nebraska
  - Weill Cornell Medicine /ID# 165887, New York, New York
  - Columbia Univ Medical Center /ID# 161934, New York, New York
  - Lenox Hill Hospital /ID# 168470, New York, New York
  - Manhattan Clinical Research, LLC /ID# 211805, New York, New York
  - DiGiovanna Institute for Medical Education & Research /ID# 171129, North Massapequa, New York
  - University of Rochester Medical Center /ID# 161664, Rochester, New York
  - Atrium Health Carolinas Medical Center /ID# 158512, Charlotte, North Carolina
  - Carolina Research /ID# 201090, Greenville, North Carolina
  - Plains Clinical Research Center, LLC /ID# 169732, Fargo, North Dakota
  - Cleveland Clinic Main Campus /ID# 209232, Cleveland, Ohio
  - The Ohio State University /ID# 164714, Columbus, Ohio
  - Optimed Research, Ltd. /ID# 167113, Columbus, Ohio
  - Great Lakes Gastroenterology Research, LLC /ID# 201777, Mentor, Ohio
  - ProMedica Physicians Digestive Healthcare /ID# 215623, Sylvania, Ohio
  - Digestive Disease Specialists /ID# 170779, Oklahoma City, Oklahoma
  - Adult Gastroenterology Associates - Gen 1 Research /ID# 208867, Tulsa, Oklahoma
  - Penn State Milton S. Hershey Medical Center /ID# 223563, Hershey, Pennsylvania
  - University of Pennsylvania /ID# 166266, Philadelphia, Pennsylvania
  - Digestive Disease Associates, LTD /ID# 232407, Wyomissing, Pennsylvania
  - Gastroenterology Associates, P.A. of Greenville /ID# 160472, Greenville, South Carolina
  - Gastro One /ID# 160418, Cordova, Tennessee
  - East Tennessee Research Institute /ID# 168747, Johnson City, Tennessee
  - Vanderbilt University Medical Center /ID# 160580, Nashville, Tennessee
  - Inquest Clinical Research /ID# 165685, Baytown, Texas
  - Texas Digestive Disease Consultants /ID# 209950, Cedar Park, Texas
  - GI Alliance /ID# 209798, Cedar Park, Texas
  - DHAT Research Institute /ID# 158226, Garland, Texas
  - Vilo Research Group Inc /ID# 207656, Houston, Texas
  - CliniCore International, LLC /ID# 158218, Houston, Texas
  - Baylor College of Medicine - Baylor Medical Center /ID# 158221, Houston, Texas
  - Precision Research Institute, LLC /ID# 201351, Houston, Texas
  - Centex Studies, Inc. - Houston /ID# 201222, Houston, Texas
  - Caprock Gastro Research, LLC /ID# 215432, Lubbock, Texas
  - Clinical Associates in Research Therapeutics of America, LLC /ID# 161376, San Antonio, Texas
  - Southern Star Research Institute, LLC /ID# 168776, San Antonio, Texas
  - Baylor Scott & White Center for Diagnostic Medicine /ID# 204130, Temple, Texas
  - Tyler Research Institute, LLC /ID# 166800, Tyler, Texas
  - Gastro Health & Nutrition - Victoria /ID# 164321, Victoria, Texas
  - Advanced Research Institute /ID# 160480, Ogden, Utah
  - Gastroenterology Consultants of Southwest Virginia /ID# 218143, Roanoke, Virginia
  - Virginia Mason Medical Center /ID# 160466, Seattle, Washington
- Argentina (5):
  - Gedyt /ID# 243423, Ciudad Autonoma de Buenos Aire, Ciuadad Autonoma de Buenos Aires
  - Cemic /Id# 167782, Ciudad Autonoma de Buenos Aire, Ciuadad Autonoma de Buenos Aires
  - Hospital Provincial del Centenario /ID# 170898, Rosario, Santa Fe Province
  - Sanatorio 9 de Julio /ID# 167780, San Miguel de Tucumán, Tucumán Province
  - Hospital Privado Univesitario /ID# 167779, Córdoba
- Austria (5):
  - Duplicate_Universitaetsklinikum St.Poelten /ID# 169048, Sankt Pölten, Lower Austria
  - Medizinische Universitaet Graz /ID# 169053, Graz, Styria
  - Ordensklinikum Linz GmbH Barmherzige Schwestern /ID# 215320, Linz, Upper Austria
  - Medizinische Universitaet Wien /ID# 169050, Vienna, Vienna
  - Landeskrankenhaus Salzburg-Universitätsklinikum der PMU (LKH) /ID# 200685, Salzburg
- Belgium (8):
  - Cliniques Universitaires de Bruxelles Hopital Erasme /ID# 200252, Brussels, Brussels Capital
  - UCL Saint-Luc /ID# 200039, Woluwe-Saint-Lambert, Brussels Capital
  - CHU UCL Namur - site Godinne /ID# 200254, Godinne, Namur
  - Universitair Ziekenhuis Leuven /ID# 170812, Leuven, Vlaams-Brabant
  - AZ-Delta /ID# 200040, Roeselare, West-Vlaanderen
  - Imelda Ziekenhuis /ID# 211100, Bonheiden
  - CHU de Liege /ID# 200253, Liège
  - Groupe Sante CHC - Clinique du MontLegia /ID# 200250, Liège
- Brazil (7):
  - Instituto Goiano de Gastroenterologia e Endoscopia Digestiva /ID# 157679, Goiânia, Goiás
  - Hospital Nossa Senhora das Graças /ID# 157671, Curitiba, Paraná
  - Hospital de Clinicas de Porto Alegre /ID# 157662, Porto Alegre, Rio Grande do Sul
  - Upeclin Fmb - Unesp /Id# 157690, Botucatu, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina de Ribeirao Preto - USP /ID# 157660, Ribeirão Preto, São Paulo
  - Faculdade de Medicina do ABC /ID# 163995, Santo André, São Paulo
  - Kaiser Clinica e Hospital Dia /ID# 157680, São José do Rio Preto, São Paulo
- Bulgaria (5):
  - UMHAT Kaspela EOOD /ID# 200797, Plovdiv
  - MHAT Hadzhi Dimitar /ID# 207945, Sliven
  - Second MHAT Sofia /ID# 200799, Sofia
  - UMHAT Sveti Ivan Rilski /ID# 210797, Sofia
  - UMHAT Tsaritsa Joanna - ISUL /ID# 209977, Sofia
- Canada (11):
  - University of Calgary /ID# 169111, Calgary, Alberta
  - Allen Whey Khye Lim Professional Corporation /ID# 169767, Edmonton, Alberta
  - Covenant Health /ID# 169114, Edmonton, Alberta
  - Fraser Clinical Trials Inc /ID# 169102, New Westminster, British Columbia
  - Percuro Clinical Research, Ltd /ID# 169109, Victoria, British Columbia
  - London Health Sciences Center- University Hospital /ID# 169103, London, Ontario
  - Scott Shulman Medicine Professional Corporation /ID# 169113, North Bay, Ontario
  - Toronto Digestive Disease Asso /ID# 169106, Vaughan, Ontario
  - Hotel Dieu de Levis /ID# 214378, Lévis, Quebec
  - CIUSSS de l'est de l'Ile-de-Montreal - Hopital Maisonneuve-Rosemont /ID# 169108, Montreal, Quebec
  - Royal Victoria Hospital / McGill University Health Centre /ID# 169104, Montreal, Quebec
- Chile (5):
  - Complejo Asistencial Dr. Sotero del Rio /ID# 169385, Santiago, Region Metropolitana Santiago
  - Servicio de Salud Occidente Hospital San Juan de Dios /ID# 171125, Santiago, Region Metropolitana Santiago
  - Servicio de Salud Araucanía Norte Hospital Victoria /ID# 213151, Victoria, Región de la Araucanía
  - Hospital Guillermo Grant Benavente de Concepción /ID# 210761, Concepción
  - Hospital Las Higueras /ID# 167093, Talcahuano
- China (25):
  - The First Affiliated Hospital of Anhui Medical University /ID# 211228, Hefei, Anhui
  - Beijing Friendship Hospital /ID# 211066, Beijing, Beijing Municipality
  - The Sixth Affiliated Hosp Sun /ID# 211231, Guangzhou, Guangdong
  - The Second Hospital of Hebei Medical University /ID# 213018, Shijiazhuang, Hebei
  - Union Hospital affiliated to Tongji Medical College of Huazhong University of Sc /ID# 211071, Wuhan, Hubei
  - Tongji Hospital Tongji Medical College of HUST /ID# 211072, Wuhan, Hubei
  - Renmin Hospital of Wuhan University /ID# 212868, Wuhan, Hubei
  - Huai'an First People's Hospital /ID# 239196, Huaian, Jiangsu
  - Nanjing Drum Tower Hospital /ID# 227439, Nanjing, Jiangsu
  - Jiangsu Province Hospital /ID# 211232, Nanjing, Jiangsu
  - Wuxi People's Hospital /ID# 218798, Wuxi, Jiangsu
  - The First Affiliated Hospital of Nanchang University /ID# 212183, Nanchang, Jiangxi
  - The First Hospital of Jilin University /ID# 212278, Changchun, Jilin
  - General Hospital of Ningxia Medical University /ID# 213911, Yinchuan, Ningxia
  - Xijing Hospital /ID# 211639, Xi'an, Shaanxi
  - Tangdu Hospital of The Fourth Military Medical University, PLA /ID# 215504, Xi'an, Shaanxi
  - Shanghai East Hospital /ID# 218791, Pudong New District, Shanghai Municipality
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine /ID# 210962, Shanghai, Shanghai Municipality
  - Renji Hospital, Shanghai Jiaotong University School of Medicine /ID# 211233, Shanghai, Shanghai Municipality
  - Shanghai General Hospital /ID# 226190, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University /ID# 211276, Chengdu, Sichuan
  - The second Affiliated hospital of Zhejiang University school of Medicine /ID# 211025, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital,Meical School Zhejiang University /ID# 211064, Hangzhou, Zhejiang
  - The Second Xiangya Hospital of Central South University /ID# 211198, Changsha
  - Shengjing Hospital of China Medical University /ID# 211646, Shenyang
- Colombia (2):
  - Oncomédica SAS /ID# 206937, Montería, Departamento de Córdoba
  - Hospital Universitario San Vic /ID# 171490, Medellín
- Croatia (5):
  - Clinical Hospital Dubrava /ID# 157475, Zagreb, City of Zagreb
  - Klinicki bolnicki centar Zagreb /ID# 157471, Zagreb, City of Zagreb
  - Klinicki bolnicki centar Zagreb /ID# 201917, Zagreb, City of Zagreb
  - Klinicki bolnicki centar Osijek /ID# 157472, Osijek, County of Osijek-Baranja
  - Klinicki bolnicki centar Split /ID# 157473, Split, Split-Dalmatia County
- Czechia (4):
  - Fakultni nemocnice u sv. Anny v Brne /ID# 239157, Brno
  - Nemocnice Ceske Budejovice a.s. /ID# 225226, České Budějovice
  - Hepato-Gastroenterologie HK, s.r.o. /ID# 163395, Hradec Králové
  - Fakultni nemocnice Ostrava /ID# 225567, Ostrava
- Denmark (4):
  - Bispebjerg and Frederiksberg Hospital /ID# 208945, Copenhagen NV, Capital Region
  - Kobenhavns Universitet - Hvidovre Hospital (HH) /ID# 202266, Hvidovre, Capital Region
  - Sjællands Universitetshospital /ID# 200033, Roskilde, Region Sjælland
  - Odense University Hospital /ID# 205602, Odense C, Region Syddanmark
- Egypt (5):
  - Clinical Research Center, Faculty of Medicine, Alexandria university. /ID# 200848, Alexandria
  - Clinical Research Center, Faculty of Medicine, Alexandria university. /ID# 226793, Alexandria
  - Clinical Research Center, Faculty of Medicine, Alexandria university. /ID# 226794, Alexandria
  - Air Force Specialized Hospital /ID# 170986, Cairo
  - National Liver Institute /ID# 171040, Menoufiya
- France (10):
  - Chu de Nice-Hopital L'Archet Ii /Id# 171577, Nice, Alpes-Maritimes
  - APHM - Hopital Nord /ID# 225825, Marseille, Bouches-du-Rhone
  - CHU Bordeaux - Hopital Haut Leveque /ID# 171579, Pessac, Gironde
  - CHU Montpellier - Hôpital Saint Eloi /ID# 223779, Montpellier, Herault
  - CHRU Nancy - Hopitaux de Brabois /ID# 200095, Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - CHU de SAINT ETIENNE - Hopital Nord /ID# 171580, Saint Priest EN Jarez, Pays de la Loire Region
  - CHU Amiens-Picardie Site Sud /ID# 171576, Amiens, Somme
  - Clinique Jules Verne /ID# 240976, Nantes
  - Hopital Beaujon /ID# 200092, Clichy, Île-de-France Region
  - Centre Médico Chirurgical Ambroise Paré Hartmann /ID# 249860, Neuilly-sur-Seine, Île-de-France Region
- Germany (20):
  - Universitaetsklinikum Freiburg /ID# 162034, Freiburg im Breisgau, Baden-Wurttemberg
  - Praxis fuer Gastroenterologie /ID# 166152, Heidelberg, Baden-Wurttemberg
  - Universitatsklinikum Mannheim /ID# 162035, Mannheim, Baden-Wurttemberg
  - Universitaetsklinikum Ulm /ID# 164992, Ulm, Baden-Wurttemberg
  - Universitaetsklinikum Erlangen /ID# 159354, Erlangen, Bavaria
  - Universitaetsklinikum Koeln /ID# 164991, Cologne, North Rhine-Westphalia
  - Praxiszentrum fuer Gastroenterologie /ID# 219069, Grevenbroich, North Rhine-Westphalia
  - Universitaetsklinikum Schleswig-Holstein Campus Kiel /ID# 159360, Kiel, Schleswig-Holstein
  - Gastroenterologische Spezialpraxis am Wittenbergplatz /ID# 219145, Berlin
  - MVZ fuer Gastroenterlogie am Bayerischen Platz /ID# 159361, Berlin
  - Charite Universitaetsklinikum Berlin - Campus Benjamin Franklin /ID# 210510, Berlin
  - DRK Kliniken Berlin Westend /ID# 166153, Berlin
  - Stadtisches Klinikum Braunschweig /ID# 163687, Braunschweig
  - Agaplesion Markus Krankenhaus /ID# 159356, Frankfurt am Main
  - Gastroenterologie Opernstrasse /ID# 163683, Kassel
  - EUGASTRO GmbH /ID# 219070, Leipzig
  - Klinikum Lueneburg /ID# 163685, Lüneburg
  - Gastroenterologische Gemeinschaftspraxis Minden /ID# 162033, Minden
  - LMU Klinikum Campus Grosshadern /ID# 210481, München
  - Universitaetsklinikum Regensburg /ID# 163686, Regensburg
- Greece (8):
  - General Hospital of Athens Ippokratio /ID# 229189, Athens, Attica
  - General Hospital of Athens Laiko /ID# 206440, Athens, Attica
  - General Hospital of Chest Diseases of Athens SOTIRIA /ID# 170915, Athens, Attica
  - Tzaneio general hospital of Piraeus /ID# 206439, Piraeus, Attica
  - University General Hospital of Heraklion PA.G.N.I /ID# 165216, Heraklion, Crete
  - General Hospital of Athens Evaggelismos and Ophthalmiatrio of Athens Polyclinic /ID# 217480, Athens
  - General Hospital of Nikaia-Piraeus "Agios Panteleimon"- general hospital dytikis /ID# 165218, Pireaus
  - Theageneio Anticancer Hospital /ID# 165217, Thessaloniki
- Israel (6):
  - Hadassah Medical Center-Hebrew University /ID# 171099, Jerusalem, Jerusalem
  - Soroka University Medical Center /ID# 171100, Beersheba, Southern District
  - The Chaim Sheba Medical Center /ID# 211278, Ramat Gan, Tel Aviv
  - Rambam Health Care Campus /ID# 171103, Haifa
  - Shaare Zedek Medical Center /ID# 163544, Jerusalem
  - Rabin Medical Center /ID# 167403, Petah Tikva
- Italy (15):
  - University of Catanzaro /ID# 200125, Catanzaro, Calabria
  - Ospedale Sant Orsola Malpighi /ID# 155611, Bologna, Emilia-Romagna
  - Ospedale Policlinico San Martino /ID# 164031, Genoa, Genova
  - Fondazione Policlinico Universitario Campus Bio-Medico di Roma /ID# 163992, Rome, Lazio
  - Azienda Ospedaliera San Camillo Forlanini /ID# 155612, Rome, Lazio
  - Azienda Ospedaliero-Universitaria Policlinico Umberto I /ID# 171226, Rome, Lazio
  - ASST Rhodense/Presidio Ospedaliero di Rho /ID# 211449, Rho, Milano
  - Istituto Clinico Humanitas /ID# 155610, Rozzano, Milano
  - Azienda Ospedaliera Universitaria Policlinico Tor Vergata /ID# 158018, Rome, Roma
  - IRCCS Ospedale Sacro Cuore Don Calabria /ID# 164041, Negrar, Verona
  - A.O. Per L'Emergenza Cannizzaro /ID# 164036, Catania
  - ASST Fatebenefratelli Sacco-Ospedale Sacco /ID# 155607, Milan
  - ASST Grande Ospedale Metropolitano Niguarda /ID# 170947, Milan
  - Azienda Ospedaliero-Universitaria di Modena /ID# 201819, Modena
  - UOC Medicina Interna e Gastroe /ID# 155608, Rome
- Japan (60):
  - Aichi Medical University Hospital /ID# 164332, Nagakute-shi, Aichi-ken
  - Daido Clinic /ID# 211479, Nagoya, Aichi-ken
  - Nagoya University Hospital /ID# 164271, Nagoya, Aichi-ken
  - Nagoya City University Hospital /ID# 164331, Nagoya, Aichi-ken
  - Fujita Health University Hospital /ID# 164261, Toyoake-shi, Aichi-ken
  - National Hospital Organization Hirosaki General Medical Center /ID# 164252, Hirosaki-shi, Aomori
  - Tokatsu Tsujinaka Hospital /ID# 164438, Abiko-shi, Chiba
  - Chiba University Hospital /ID# 209632, Chiba, Chiba
  - Tsujinaka Hospital Kashiwanoha /ID# 208964, Kashiwa-shi, Chiba
  - Toho University Sakura Medical Center /ID# 164254, Sakura-shi, Chiba
  - Fukuoka University Chikushi Hospital /ID# 209055, Chikushino-shi, Fukuoka
  - Saiseikai Fukuoka Genaral Hospital /ID# 225639, Fukuoka, Fukuoka
  - Fukuoka University Hospital /ID# 226189, Fukuoka, Fukuoka
  - Kurume University Hospital /ID# 164427, Kurume-shi, Fukuoka
  - Gifu University Hospital /ID# 208081, Gifu, Gifu
  - Ogaki Municipal Hospital /ID# 226010, Ogaki-shi, Gifu
  - National Hospital Organization Takasaki General Medical Center /ID# 164437, Takasaki-shi, Gunma
  - NHO Fukuyama Medical Center /ID# 164439, Fukuyama-shi, Hiroshima
  - Hiroshima University Hospital /ID# 164426, Hiroshima, Hiroshima
  - Asahikawa Medical University Hospital /ID# 164433, Asahikawa-shi, Hokkaido
  - Hokkaido P.W.F.A.C. Sapporo-Kosei General Hospital /ID# 164251, Sapporo, Hokkaido
  - Sapporo Medical University Hospital /ID# 164432, Sapporo, Hokkaido
  - Sapporo IBD Clinic /ID# 225923, Sapporo, Hokkaido
  - Sapporo Higashi Tokushukai Hospital /ID# 208488, Sapporo, Hokkaido
  - Aoyama Clinic /ID# 164425, Kobe, Hyōgo
  - Hyogo Medical University Hospital /ID# 164424, Nishinomiya-shi, Hyōgo
  - Kanazawa University Hospital /ID# 169224, Kanazawa, Ishikawa-ken
  - Sameshima Hospital /ID# 211181, Kagoshima, Kagoshima-ken
  - Tokai University Hospital /ID# 209204, Isehara-shi, Kanagawa
  - Gokeikai Ofuna Chuo Hospital /ID# 169300, Kamakura-shi, Kanagawa
  - St. Marianna University Hospital /ID# 226728, Kawasaki-shi, Kanagawa
  - Kitasato University Hospital /ID# 169226, Sagamihara-shi, Kanagawa
  - Colo-proctology Center Matsushima Clinic /ID# 225914, Yokohama, Kanagawa
  - Showa University Fujigaoka Hospital /ID# 209555, Yokohama, Kanagawa
  - Mie University Hospital /ID# 203633, Tsu, Mie-ken
  - Yokkaichi Hazu Medical Center /ID# 164441, Yokkaichi-shi, Mie-ken
  - Tohoku University Hospital /ID# 164430, Sendai, Miyagi
  - Nagasaki University Hospital /ID# 202674, Nagasaki, Nagasaki
  - Nara Medical University Hospital /ID# 169225, Kashihara-shi, Nara
  - Kinshukai Infusion Clinic /ID# 226747, Osaka, Osaka
  - Osaka Medical and Pharmaceutical University Hospital /ID# 226035, Takatsuki-shi, Osaka
  - Saga University Hospital /ID# 209396, Saga, Saga-ken
  - Tokitokai Tokito clinic /ID# 164253, Saitama-shi, Saitama
  - Shiga University of Medical Science Hospital /ID# 164440, Ōtsu, Shiga
  - Hamamatsu University Hospital /ID# 226727, Hamamatsu, Shizuoka
  - Matsuda Hospital /ID# 226616, Hamamatsu, Shizuoka
  - NHO Shizuoka Medical Center /ID# 164435, Sunto-gun, Shizuoka
  - Tokyo Medical And Dental University Hospital /ID# 164258, Bunkyo-ku, Tokyo
  - St.Luke's International Hospital /ID# 225822, Chuo-ku, Tokyo
  - Tokai University Hachioji Hospital /ID# 226899, Hachioji-shi, Tokyo
  - Teikyo University Hospital /ID# 225588, Itabashi-ku, Tokyo
  - The Jikei University Hospital /ID# 164434, Minato-ku, Tokyo
  - Kitasato University Kitasato Institute Hospital /ID# 164256, Minato-ku, Tokyo
  - Kyorin University Hospital /ID# 164259, Mitaka-shi, Tokyo
  - NTT Medical Center Tokyo /ID# 225587, Shinagawa-ku, Tokyo
  - Keio University Hospital /ID# 203629, Shinjuku-ku, Tokyo
  - Japanese Red Cross Wakayama Medical Center /ID# 171195, Wakayama, Wakayama
  - Wakayama Medical University Hospital /ID# 169487, Wakayama, Wakayama
  - Yamagata University Hospital /ID# 171474, Yamagata, Yamagata
  - Tokuyama Central Hospital /ID# 226011, Shunan-shi, Yamaguchi
- Latvia (2):
  - VCA Polyclinic Aura /ID# 163802, Riga
  - Pauls Stradins Clinical University Hospital /ID# 163803, Riga
- Lithuania (2):
  - Hospital of Lithuanian University of Health Sciences Kaunas Clinics /ID# 170714, Kaunas
  - Vilnius University Hospital Santaros Klinikos /ID# 170614, Vilnius
- Universiti Sains Malaysia /ID# 221971, Kelantan, Kelantan, Malaysia
- Mexico (3):
  - JM Research SC /ID# 203593, Cuernavaca, Morelos
  - Unidad de Atencion Medica e Investigacion en Salud /ID# 203595, Mérida, Yucatán
  - Health Pharma Professional Research S.A de C.V /ID# 203597, Del. Benito Juárez
- Netherlands (2):
  - Academisch Medisch Centrum /ID# 157959, Amsterdam
  - Elisabeth Tweesteden Ziekenhuis /ID# 163767, Tilburg
- New Zealand (6):
  - Tauranga Hospital /ID# 212792, Tauranga South, Bay of Plenty
  - Christchurch Hospital /ID# 205342, Christchurch, Canterbury
  - Dunedin Hospital /ID# 212790, Otago, Otago
  - Waikato Hospital /ID# 212789, Hamilton, Waikato Region
  - Wellington Regional Hospital /ID# 205343, Newtown, Wellington Region
  - Hutt Hospital /ID# 212786, Lower Hutt
- Poland (12):
  - Vitamed Gałaj i Cichomski Sp.j. /ID# 213283, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Gastromed Sp. z o.o /ID# 230978, Torun, Kuyavian-Pomeranian Voivodeship
  - Centrum Medyczne Plejady /ID# 170633, Krakow, Lesser Poland Voivodeship
  - Vistamed /ID# 210105, Wroclaw, Lower Silesian Voivodeship
  - Centrum Zdrowia MDM /ID# 170597, Warsaw, Masovian Voivodeship
  - WIP Warsaw IBD Point Profesor Kierkus /ID# 216102, Warsaw, Masovian Voivodeship
  - Panstwowy Instytut Medyczny MSWiA w Warszawie /ID# 170601, Warsaw, Masovian Voivodeship
  - Narodowy Instytut Onkologii im. Marii Skłodowskiej-Curie Panstwowy Instytut Bada /ID# 170600, Warsaw, Masovian Voivodeship
  - NZOZ Vivamed Jadwiga Miecz /ID# 216307, Warsaw, Masovian Voivodeship
  - Endoskopia Sp. z o.o. /ID# 170598, Sopot, Pomeranian Voivodeship
  - NZOZ All-Medicus /ID# 170596, Katowice, Silesian Voivodeship
  - H-T. Centrum Medyczne - Endoterapia /ID# 230979, Tychy, Silesian Voivodeship
- Portugal (8):
  - Hospital da Senhora da Oliveira Guimaraes, EPE /ID# 165580, Guimarães, Braga District
  - Centro Hospitalar Universitário do Algarve, EPE - Hospital de Portimão /ID# 166551, Portimão, Faro District
  - Centro Hospitalar de Entre Douro e Vouga /ID# 166052, Santa Maria DA Feira, Porto District
  - Hospital Garcia de Orta, EPE /ID# 165583, Almada
  - Centro Hospitalar e Universitario de Coimbra, EPE /ID# 166054, Coimbra
  - Centro Hospitalar Universitario Lisboa Central, EPE - Hospital dos Capuchos /ID# 165582, Lisbon
  - Centro Hospitalar Universitario de Sao Joao, EPE /ID# 165581, Porto
  - Centro Hosp de Tondela-Viseu /ID# 166053, Viseu
- Puerto Rico (3):
  - Ponce Medical School Foundation /ID# 221244, Ponce
  - San Jorge Children Hospital /ID# 166954, San Juan
  - VA Caribbean Healthcare System /ID# 221245, San Juan
- Romania (6):
  - Clinica GASTRO MED SRL /ID# 224169, Cluj-Napoca, Cluj
  - Sana Monitoring /Id# 224166, Bucharest
  - Fundeni Clinical Institute /ID# 171264, Bucharest
  - Fundeni Clinical Institute /ID# 224168, Bucharest
  - Cabinet Particular Policlinic Algomed /ID# 171266, Timișoara
  - Duplicate_Centrul Medical Tuculanu SRL /ID# 171268, Timișoara
- Russia (17):
  - Interdisctrict Multidisciplinary Hospital /ID# 203335, Anzorey, Kabardino-Balkarskaya Respublika
  - GBUZ Allergology and Immunology Center of Ministry of Health of Kabardino-Bal /ID# 233973, Nal'chik, Kabardino-Balkarskaya Respublika
  - Immanuel Kant Baltic Federal University /ID# 204888, Kaliningrad, Kaliningrad Oblast
  - Kuzbass Regional Clinical Hospital /ID# 165750, Kemerovo, Kemerovo Oblast
  - Uninova Medical Center /ID# 229216, Saint Petersburg, Leningradskaya Oblast'
  - Arsvita Clinic /ID# 208946, Korolyov, Moscow Oblast
  - Perm Clinical Center of the Federal Medical and Biological Agency /ID# 227457, Perm, Permskiy Kray
  - City Clinical Hospital #40 /ID# 203370, Sestroretsk, Sankt-Peterburg
  - Regional Clinical Hospital #1 /ID# 165754, Tyumen, Tyumen Oblast
  - Clinic of New Technologies of Medicine /ID# 203369, Dzerzhinskiy
  - First Moscow State Medical University n.a I.M. Sechenov /ID# 204978, Moscow
  - National Medical Research Center of Coloproctology n.a. A. N. Ryzhikh /ID# 203512, Moscow
  - Central Clinical Hospital RZHD Medicine /ID# 204917, Moscow
  - Novosibirski Gastrocenter /ID# 229855, Novosibirsk
  - Euromedservice /ID# 204892, Pushkin
  - International Medical Center SOGAZ /ID# 206727, Saint Petersburg
  - Ulyanovsk Regional Clinical Hospital /ID# 203368, Ulyanovsk
- Serbia (6):
  - Clinical Hosp Center Zvezdara /ID# 200151, Belgrade, Beograd
  - University Clinical Center Serbia /ID# 200152, Belgrade, Beograd
  - Clin Hosp Ctr Bezanijska Kosa /ID# 202059, Belgrade, Beograd
  - Clinical Center Vojvodina /ID# 156910, Novi Sad, Vojvodina
  - Clinical Hospital Center Dr Dragisa Misovic - Dedinje /ID# 224926, Belgrade
  - General Hospital Leskovac /ID# 207226, Leskovac
- KL Ling Gastroenterology and Liver Clinic /ID# 205738, Singapore, Singapore
- Slovakia (4):
  - Fakultna nemocnica s poliklinikou F.D. Roosevelta Banska Bystrica /ID# 164347, Banská Bystrica
  - KM Management, spol. s.r.o. /ID# 206602, Nitra
  - Fakultna nemocnica s poliklinikou Nove Zamky /ID# 224099, Nové Zámky
  - GASTRO I., s.r.o. /ID# 164346, Prešov
- Univ Medical Ctr Ljubljana /ID# 210627, Ljubljana, Slovenia
- South Africa (6):
  - Farmovs (Pty) Ltd /Id# 207537, Bloemfontein, Free State
  - Clinresco Centers /ID# 239824, Johannesburg, Gauteng
  - Allergy & Immunology (AIU) /ID# 171441, Cape Town, Western Cape
  - Dr JP Wright /ID# 171138, Cape Town, Western Cape
  - Private Practice Dr MN Rajabally /ID# 171137, Cape Town, Western Cape
  - Spoke Research Inc /ID# 229905, CAPE TOWN Milnerton, Western Cape
- South Korea (11):
  - Hanyang University Gurihospital /ID# 158702, Guri-si, Gyeonggido
  - CHA University Bundang Medical Center /ID# 158710, Seongnam-si, Gyeonggido
  - The Catholic University of Korea, ST. Vincent's Hospital /ID# 158706, Suwon, Gyeonggido
  - Kangbuk Samsung Hospital /ID# 158707, Seoul, Seoul Teugbyeolsi
  - Yonsei University Health System Severance Hospital /ID# 158701, Seoul, Seoul Teugbyeolsi
  - Inje University Haeundae Hospital /ID# 203028, Busan
  - Dong-A University Hospital /ID# 158705, Busan
  - Pusan National University Hospital /ID# 158711, Busan
  - Yeungnam University Medical Center /ID# 158703, Daegu
  - The Catholic University of Korea, Daejeon St.Mary's Hospital /ID# 242378, Daejeon
  - Samsung Medical Center /ID# 158704, Seoul
- Spain (12):
  - Hospital Arquitecto Marcide - Complejo Hospitalario Universitario de Ferrol /ID# 159440, Ferrol, A Coruna
  - Consorci Corporacio Sanitaria Parc Tauli Sabadell /ID# 159461, Sabadell, Barcelona
  - Hospital Universitario Puerta de Hierro, Majadahonda /ID# 159443, Majadahonda, Madrid
  - Hospital Alvaro Cunqueiro CHUVI /ID# 167360, Vigo, Pontevedra
  - Hospital de Cabuenes /ID# 170748, Gijón, Principality of Asturias
  - Hospital Clinic de Barcelona /ID# 159439, Barcelona
  - Hospital Universitario Reina Sofia /ID# 167058, Córdoba
  - Hospital Universitario La Paz /ID# 159459, Madrid
  - Complejo Hospitalario Universitario de Pontevedra /ID# 216182, Pontevedra
  - Hospital Universitario de Salamanca /ID# 159446, Salamanca
  - Hospital Universitario Virgen Macarena /ID# 159968, Seville
  - Hospital Universitario Miguel Servet /ID# 159445, Zaragoza
- Sweden (3):
  - Alingsas lasarett /ID# 202074, Alingsås, Västra Götaland County
  - Sahlgrenska University Hospital Molndal /ID# 202843, Mölndal, Västra Götaland County
  - Danderyds sjukhus AB /ID# 202035, Stockholm
- Switzerland (2):
  - Universitatsspital Zurich /ID# 202910, Zurich, Canton of Zurich
  - Inselspital, Universitätsspital Bern /ID# 202911, Bern
- Taiwan (6):
  - Chung Shan Medical University Hospital /ID# 163651, Taichung
  - China Medical University Hospital /ID# 160189, Taichung
  - Taichung Veterans General Hospital /ID# 163649, Taichung
  - National Taiwan University Hospital /ID# 162187, Taipei
  - Taipei Veterans General Hosp /ID# 163650, Taipei
  - Linkou Chang Gung Memorial Hospital /ID# 222877, Taoyuan
- Turkey (Türkiye) (9):
  - Acibadem Kozyatagi Hospital /ID# 213276, Kadıköy, Istanbul
  - Erciyes University Medical Fac /ID# 171291, Melikgazi, Kayseri
  - Ankara Univ Medical Faculty /ID# 167210, Ankara
  - Inonu Universitesi Turgut Ozal /ID# 203981, Battalgazi/malatya
  - Uludag University Medical Faculty /ID# 204182, Bursa
  - Fırat University Medical Facul /ID# 171292, Elâzığ
  - Istanbul University-Cerrahpasa, Cerrahpasa Medical Faculty /ID# 167207, Istanbul
  - Marmara Universitesi Pendik Egitim ve Arastirma Hastanesi /ID# 171293, Istanbul
  - Sisli Etfal Train & Res Hosp /ID# 171409, Şişli
- Ukraine (5):
  - CNE Regional Clinical Hospital of Ivano-Frankivsk RC /ID# 203367, Ivano-Frankivsk
  - Municipal Nonprofit Enterprise Kherson city clinical hospital n.a. Y.Y. Karabel /ID# 224350, Kherson
  - Kyiv Municipal Clinical Hospital #18 /ID# 224348, Kyiv
  - Medical Center "OK!Clinic+" /ID# 205482, Kyiv
  - CNPE of Kyiv Regional Council Kyiv Regional Hospital /ID# 224343, Kyiv
- United Kingdom (10):
  - Royal Devon University Healthcare NHS Foundation Trust /ID# 157587, Exeter, Devon
  - University Hospital Southampton NHS Foundation Trust /ID# 210813, Southampton, Hampshire
  - Barts Health NHS Trust /ID# 157590, London, London, City of
  - Barnsley Hospital NHS Foundation Trust /ID# 202770, Barnsley
  - Cambridge University Hospitals NHS Foundation Trust /ID# 158040, Cambridge
  - NHS Lothian /ID# 208802, Edinburgh
  - Liverpool University Hospitals NHS Foundation Trust /ID# 203858, Liverpool
  - King's College Hospital NHS Foundation Trust /ID# 158766, London
  - The Newcastle Upon Tyne Hospitals NHS Foundation Trust /ID# 158041, Newcastle upon Tyne
  - St George's University Hospitals NHS Foundation Trust /ID# 208378, Tooting

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Panaccione R, Melmed GY, Drobne D, Kaur M, Danese S, Hisamatsu T, Kalabic J, Chen S, Cheng L, Duan WR, Shah S, Louis E. Impact of Extended Risankizumab Treatment in Patients With Ulcerative Colitis Who Did Not Respond to Induction Treatment. Clin Gastroenterol Hepatol. 2025 Sep 13:S1542-3565(25)00797-9. doi: 10.1016/j.cgh.2025.09.007. Online ahead of print. PMID 40953785
- [Derived] Reinisch W, Loftus EV Jr, Schreiber S, Rubin DT, Louis E, Hecht PM, Barrachina EM, Kalabic J, Vladea R, Sharma D, Duan WR, Zhang Y, Panaccione R. Corticosteroid-sparing effects of risankizumab efficacy and safety in patients with moderately to severely active ulcerative colitis. J Crohns Colitis. 2025 Apr 4;19(4):jjaf025. doi: 10.1093/ecco-jcc/jjaf025. PMID 40168091
- [Derived] Panaccione R, Louis E, Colombel JF, D'Haens G, Peyrin-Biroulet L, Dubinsky M, Takeuchi K, Rubin DT, Kalabic J, Chien KB, Chen S, Cheng L, Zhang Y, Duan WR, Vladea R, Hecht PM, Morisset P, Schreiber S, Ferrante M. Risankizumab efficacy and safety based on prior inadequate response or intolerance to advanced therapy: post hoc analysis of the INSPIRE and COMMAND phase 3 studies. J Crohns Colitis. 2025 Jan 11;19(1):jjaf005. doi: 10.1093/ecco-jcc/jjaf005. PMID 39804294
- [Derived] Louis E, Schreiber S, Panaccione R, Bossuyt P, Biedermann L, Colombel JF, Parkes G, Peyrin-Biroulet L, D'Haens G, Hisamatsu T, Siegmund B, Wu K, Boland BS, Melmed GY, Armuzzi A, Levine P, Kalabic J, Chen S, Cheng L, Shu L, Duan WR, Pivorunas V, Sanchez Gonzalez Y, D'Cunha R, Neimark E, Wallace K, Atreya R, Ferrante M, Loftus EV Jr; INSPIRE and COMMAND Study Group. Risankizumab for Ulcerative Colitis: Two Randomized Clinical Trials. JAMA. 2024 Sep 17;332(11):881-897. doi: 10.1001/jama.2024.12414. PMID 39037800
- See also: Related Info — https://www.abbvieclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was comprised of 2 SubStudies, each had 2 Periods.
Period: Substudy 1 Period 1
Arm/Group | Substudy 1, Induction Period 1: Double-blind Placebo IV | Substudy 1, Induction Period 1: Double-blind Risankizumab 600mg IV | Substudy 1, Induction Period 1: Double-blind Risankizumab 1200mg IV | Substudy 1, Induction Period 1: Double-blind Risankizumab 1800mg IV | Substudy 1, Induction Period 1: Open-label Risankizumab 1800mg IV | Substudy 1, Induction Period 2: Double-blind Risankizumab 180mg SC | Substudy 1, Induction Period 2: Double-blind Risankizumab 360mg SC | Substudy 1, Induction Period 2: Double-blind Risankizumab 1800mg IV | Substudy 1, Induction Period 2: Double-blind Risankizumab 1800mg IV Pbo | Substudy 2, Induction Period 1: Double-blind Placebo IV | Substudy 2, Induction Period 1: Double-blind Risankizumab 1200mg IV | Substudy 2, Induction Period 2: Double-blind Risankizumab 180mg SC | Substudy 2, Induction Period 2: Double-blind Risankizumab 360mg SC | Substudy 2, Induction Period 2: Double-blind Risankizumab 1200mg IV | Substudy 2, Induction Period 2: Double-blind Risankizumab 1200mg IV Pbo
Started | 60 | 61 | 61 | 58 | 341 (341 enrolled, 340 treated) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 53 | 55 | 58 | 57 | 306 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 7 | 6 | 3 | 1 | 35 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 5 | 2 | 2 | 0 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — WITHDREW CONSENT | 1 | 2 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 1 | 1 | 0 | 20 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Enrolled but not Treated | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Substudy 1 Period 2
Arm/Group | Substudy 1, Induction Period 1: Double-blind Placebo IV | Substudy 1, Induction Period 1: Double-blind Risankizumab 600mg IV | Substudy 1, Induction Period 1: Double-blind Risankizumab 1200mg IV | Substudy 1, Induction Period 1: Double-blind Risankizumab 1800mg IV | Substudy 1, Induction Period 1: Open-label Risankizumab 1800mg IV | Substudy 1, Induction Period 2: Double-blind Risankizumab 180mg SC | Substudy 1, Induction Period 2: Double-blind Risankizumab 360mg SC | Substudy 1, Induction Period 2: Double-blind Risankizumab 1800mg IV | Substudy 1, Induction Period 2: Double-blind Risankizumab 1800mg IV Pbo | Substudy 2, Induction Period 1: Double-blind Placebo IV | Substudy 2, Induction Period 1: Double-blind Risankizumab 1200mg IV | Substudy 2, Induction Period 2: Double-blind Risankizumab 180mg SC | Substudy 2, Induction Period 2: Double-blind Risankizumab 360mg SC | Substudy 2, Induction Period 2: Double-blind Risankizumab 1200mg IV | Substudy 2, Induction Period 2: Double-blind Risankizumab 1200mg IV Pbo
Started | 0 | 0 | 0 | 0 | 0 | 72 | 70 (70 enrolled, 69 treated) | 36 | 37 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 65 | 57 | 34 | 35 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 7 | 13 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — WITHDREW CONSENT | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 5 | 5 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — COVID-19 LOGISTICAL RESTRICTIONS | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Enrolled but not Treated | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Substudy 2 Period 1
Arm/Group | Substudy 1, Induction Period 1: Double-blind Placebo IV | Substudy 1, Induction Period 1: Double-blind Risankizumab 600mg IV | Substudy 1, Induction Period 1: Double-blind Risankizumab 1200mg IV | Substudy 1, Induction Period 1: Double-blind Risankizumab 1800mg IV | Substudy 1, Induction Period 1: Open-label Risankizumab 1800mg IV | Substudy 1, Induction Period 2: Double-blind Risankizumab 180mg SC | Substudy 1, Induction Period 2: Double-blind Risankizumab 360mg SC | Substudy 1, Induction Period 2: Double-blind Risankizumab 1800mg IV | Substudy 1, Induction Period 2: Double-blind Risankizumab 1800mg IV Pbo | Substudy 2, Induction Period 1: Double-blind Placebo IV | Substudy 2, Induction Period 1: Double-blind Risankizumab 1200mg IV | Substudy 2, Induction Period 2: Double-blind Risankizumab 180mg SC | Substudy 2, Induction Period 2: Double-blind Risankizumab 360mg SC | Substudy 2, Induction Period 2: Double-blind Risankizumab 1200mg IV | Substudy 2, Induction Period 2: Double-blind Risankizumab 1200mg IV Pbo
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 325 | 652 (652 enrolled, 650 treated.) | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 297 | 637 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 28 | 15 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 2 | 0 | 0 | 0 | 0
Not completed — WITHDREW CONSENT | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 4 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 1 | 0 | 0 | 0 | 0
Not completed — COVID-19 INFECTION | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — COVID-19 LOGISTICAL RESTRICTIONS | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4 | 0 | 0 | 0 | 0
Not completed — Enrolled but not Treated | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Period: Substudy 2 Period 2
Arm/Group | Substudy 1, Induction Period 1: Double-blind Placebo IV | Substudy 1, Induction Period 1: Double-blind Risankizumab 600mg IV | Substudy 1, Induction Period 1: Double-blind Risankizumab 1200mg IV | Substudy 1, Induction Period 1: Double-blind Risankizumab 1800mg IV | Substudy 1, Induction Period 1: Open-label Risankizumab 1800mg IV | Substudy 1, Induction Period 2: Double-blind Risankizumab 180mg SC | Substudy 1, Induction Period 2: Double-blind Risankizumab 360mg SC | Substudy 1, Induction Period 2: Double-blind Risankizumab 1800mg IV | Substudy 1, Induction Period 2: Double-blind Risankizumab 1800mg IV Pbo | Substudy 2, Induction Period 1: Double-blind Placebo IV | Substudy 2, Induction Period 1: Double-blind Risankizumab 1200mg IV | Substudy 2, Induction Period 2: Double-blind Risankizumab 180mg SC | Substudy 2, Induction Period 2: Double-blind Risankizumab 360mg SC | Substudy 2, Induction Period 2: Double-blind Risankizumab 1200mg IV | Substudy 2, Induction Period 2: Double-blind Risankizumab 1200mg IV Pbo
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 71 | 71 (71 enrolled; 70 treated) | 68 | 174 (174 enrolled; 173 treated)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 65 | 65 | 61 | 164
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 7 | 10
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Not completed — WITHDREW CONSENT | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 2 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 3 | 4
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Enrolled but not Treated | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Includes all enrolled subjects that received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Substudy 1, Induction Period 1: Double-blind Placebo IV | Substudy 1, Induction Period 1: Double-blind Risankizumab 600mg IV | Substudy 1, Induction Period 1: Double-blind Risankizumab 1200mg IV | Substudy 1, Induction Period 1: Double-blind Risankizumab 1800mg IV | Substudy 1, Induction Period 1: Open-label Risankizumab 1800mg IV | Substudy 2, Induction Period 1: Double-blind Placebo IV | Substudy 2, Induction Period 1: Double-blind Risankizumab 1200mg IV | Total
Number analyzed (Participants) | 60 | 61 | 61 | 58 | 340 | 325 | 650 | 1555
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Population includes subjects who received at least one dose of study drug.
  years
    Substudy 1: number analyzed (Participants) | 60 | 61 | 61 | 58 | 340 | 0 | 0 | 580
    Substudy 1 | 44.4 (14.09) | 43.0 (14.90) | 41.8 (13.80) | 40.9 (13.73) | 40.4 (14.17) |  |  | 42.5 (14.12)
    Substudy 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 325 | 650 | 975
    Substudy 2 |  |  |  |  |  | 42.8 (14.30) | 41.8 (13.47) | 42.1 (13.75)
Age, Customized [Count of Participants; unit: Participants]
  Age Group: 18 - <40 | 25 | 27 | 30 | 33 | 175 | 147 | 313 | 750
  Age Group: 40 - <65 | 29 | 27 | 27 | 20 | 143 | 153 | 299 | 698
  Age Group: ≥65 | 6 | 7 | 4 | 5 | 22 | 25 | 38 | 107
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 21 | 26 | 27 | 145 | 124 | 265 | 632
  Male | 36 | 40 | 35 | 31 | 195 | 201 | 385 | 923
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 6 | 1 | 21 | 20 | 44 | 97
  Not Hispanic or Latino | 57 | 59 | 55 | 57 | 319 | 305 | 606 | 1458
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Asian | 14 | 11 | 15 | 11 | 47 | 96 | 171 | 365
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 1 | 2 | 3 | 7 | 12 | 28
  White | 44 | 49 | 45 | 45 | 290 | 218 | 461 | 1152
  More than one race | 0 | 0 | 0 | 0 | 0 | 4 | 5 | 9
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Adapted Mayo Score [Mean (Standard Deviation); unit: Adapted Mayo Score 0 - 9] — The Adapted Mayo Score is a composite score of UC disease activity based on the following 3 subscores:
  1. Stool frequency subscore (SFS), scored from 0 (normal number of stools) to 3 (5 or more stools more than normal)
  2. Rectal bleeding subscore (RBS), scored from 0 (no blood seen) to 3 (blood alone passed)
  3. Endoscopic subscore, scored from 0 (normal or inactive disease) to 3 (severe disease, spontaneous bleeding, ulceration) The overall Adapted Mayo score ranges from 0 to 9 where higher scores represent more severe disease. Population: Population includes subjects who received at least one dose of study drug and had available data for analysis.
  Adapted Mayo Score 0 - 9
    Substudy 1 - ITT1A Population: number analyzed (Participants) | 60 | 61 | 61 | 58 | 0 | 0 | 0 | 240
    Substudy 1 - ITT1A Population | 7.012 (1.1645) | 6.929 (1.2240) | 7.011 (1.1288) | 7.150 (1.3908) |  |  |  | 7.024 (1.2240)
    Substudy 1 - ITT1B Population: number analyzed (Participants) | 0 | 0 | 0 | 0 | 340 | 0 | 0 | 340
    Substudy 1 - ITT1B Population |  |  |  |  | 7.179 (1.2279) |  |  | 7.179 (1.2279)
    Substudy 2 - ITT2 Population: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 325 | 649 | 974
    Substudy 2 - ITT2 Population |  |  |  |  |  | 7.052 (1.2800) | 7.068 (1.2173) | 7.063 (1.2380)

OUTCOME MEASURES:

1. Primary Outcome: Sub-Study 1: Percentage of Participants Achieving Clinical Remission Per Adapted Mayo Score
Description: The Adapted Mayo Score is a composite score of UC disease activity based on the following 3 subscores:
  1. Stool frequency subscore (SFS), scored from 0 (normal number of stools) to 3 (5 or more stools more than normal)
  2. Rectal bleeding subscore (RBS), scored from 0 (no blood seen) to 3 (blood alone passed)
  3. Endoscopic subscore, scored from 0 (normal or inactive disease) to 3 (severe disease, spontaneous bleeding, ulceration)
  The overall Adapted Mayo score ranges from 0 to 9 where higher scores represent more severe disease.
  For Sub-Study 1, clinical remission was defined as SFS ≤ 1, and not greater than baseline, RBS of 0, and endoscopic subscore ≤ 1.
Time Frame: Week 12
Population: ITT1A includes all randomized subjects who received at least one dose of study drug during Induction Period 1 from Substudy 1.
  ITT1B includes all the additional subjects who received at least one dose of risankizumab 1800 mg IV treatment group after 240 subjects were randomized during Induction Period 1 from Substudy 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Substudy 1, Induction Period 1: Double-blind Placebo IV | Substudy 1, Induction Period 1: Double-blind Risankizumab 600mg IV | Substudy 1, Induction Period 1: Double-blind Risankizumab 1200mg IV | Substudy 1, Induction Period 1: Double-blind Risankizumab 1800mg IV | Substudy 1, Induction Period 1: Open-label Risankizumab 1800mg IV
Number analyzed (Participants) | 60 | 61 | 61 | 58 | 340
Participants | 1 | 7 | 6 | 6 | 42
Statistical Analysis 1: Comparison: Substudy 1, Induction Period 1: Double-blind Placebo IV vs Substudy 1, Induction Period 1: Double-blind Risankizumab 600mg IV; Test type: Superiority; p = 0.0324, Cochran-Mantel-Haenszel — P-value ≤ 0.05; Based on Cochran-Mantel-Haenszel (CMH) test stratified by baseline corticosteroid use (yes, no) and baseline adapted mayo score (≤ 7, > 7); Adjusted Risk Difference = 9.6, 90% CI 2-sided [2.2 to 17.0] — Risk difference = (risankizumab - Placebo)
Statistical Analysis 2: Comparison: Substudy 1, Induction Period 1: Double-blind Placebo IV vs Substudy 1, Induction Period 1: Double-blind Risankizumab 1200mg IV; Test type: Superiority; p = 0.0460, Cochran-Mantel-Haenszel — P-value ≤ 0.05; [statistical method as in outcome 1, analysis 1]; Adjusted Risk Difference = 8.4, 90% CI 2-sided [1.5 to 15.3] — Risk difference = (risankizumab - Placebo)
Statistical Analysis 3: Comparison: Substudy 1, Induction Period 1: Double-blind Placebo IV vs Substudy 1, Induction Period 1: Double-blind Risankizumab 1800mg IV; Test type: Superiority; p = 0.0397, Cochran-Mantel-Haenszel — P-value ≤ 0.05; [statistical method as in outcome 1, analysis 1]; Adjusted Risk Difference = 8.7, 90% CI 2-sided [1.7 to 15.6] — Risk difference = (risankizumab - Placebo)

2. Primary Outcome: Sub-Study 2: Percentage of Participants Achieving Clinical Remission Per Adapted Mayo Score
Description: The Adapted Mayo Score is a composite score of UC disease activity based on the following 3 subscores:
  1. Stool frequency subscore (SFS), scored from 0 (normal number of stools) to 3 (5 or more stools more than normal)
  2. Rectal bleeding subscore (RBS), scored from 0 (no blood seen) to 3 (blood alone passed)
  3. Endoscopic subscore, scored from 0 (normal or inactive disease) to 3 (severe disease, spontaneous bleeding, ulceration)
  The overall Adapted Mayo score ranges from 0 to 9 where higher scores represent more severe disease.
  For Sub-Study 2, clinical remission was defined as SFS ≤ 1, and not greater than baseline, RBS of 0, and endoscopic subscore ≤ 1. Evidence of friability during endoscopy in subjects with otherwise "mild" endoscopic activity will confer an endoscopic subscore of 2.
Time Frame: Week 12
Population: ITT2 population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Substudy 2, Induction Period 1: Double-blind Placebo IV | Substudy 2, Induction Period 1: Double-blind Risankizumab 1200mg IV
Number analyzed (Participants) | 325 | 650
percentage of participants | 6.2 [3.6 to 8.9] | 20.3 [17.2 to 23.4]
Statistical Analysis 1: Comparison: Substudy 2, Induction Period 1: Double-blind Placebo IV vs Substudy 2, Induction Period 1: Double-blind Risankizumab 1200mg IV; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Type I error rate control; Stratified by Advanced Therapy-IR status (yes vs no), Baseline steroid use (yes vs. no) and Baseline Adapted Mayo Score (≤ 7, > 7); Adjusted Risk Difference = 14.0, 95% CI 2-sided [10.0 to 18.0]

3. Secondary Outcome: Sub-Study 1: Percentage of Participants Achieving Endoscopic Improvement
Description: Endoscopic improvement is defined as endoscopy subscore of 0 or 1.
  Endoscopies were assessed by a blinded central reader and scored according to the following scale: 0 = Normal or inactive disease; 1 = Mild disease (erythema, decreased vascular pattern); 2 = Moderate disease (marked erythema, lack of vascular pattern, any friability, erosions); 3 = Severe disease (spontaneous bleeding, ulceration).
Time Frame: Week 12
Population: Includes ITT1A and ITT1B populations.
Measure: Count of Participants; unit: Participants
Arm/Group | Substudy 1, Induction Period 1: Double-blind Placebo IV | Substudy 1, Induction Period 1: Double-blind Risankizumab 600mg IV | Substudy 1, Induction Period 1: Double-blind Risankizumab 1200mg IV | Substudy 1, Induction Period 1: Double-blind Risankizumab 1800mg IV | Substudy 1, Induction Period 1: Open-label Risankizumab 1800mg IV
Number analyzed (Participants) | 60 | 61 | 61 | 58 | 340
Participants | 3 | 15 | 8 | 9 | 61
Statistical Analysis 1: Comparison: Substudy 1, Induction Period 1: Double-blind Placebo IV vs Substudy 1, Induction Period 1: Double-blind Risankizumab 600mg IV; Test type: Superiority; p = 0.0028, Cochran-Mantel-Haenszel — P-value ≤ 0.01; Stratified by baseline corticosteroid use (yes, no) and baseline adapted mayo score (<= 7, > 7); Adjusted Risk Difference = 18.7, 90% CI 2-sided [8.4 to 29.0] — Risk difference = (risankizumab - Placebo)
Statistical Analysis 2: Comparison: Substudy 1, Induction Period 1: Double-blind Placebo IV vs Substudy 1, Induction Period 1: Double-blind Risankizumab 1200mg IV; Test type: Superiority; p = 0.0968, Cochran-Mantel-Haenszel — P-value ≤ 0.1; Stratified by baseline corticosteroid use (yes, no) and baseline adapted mayo score (<= 7, > 7); Adjusted Risk Difference = 8.4, 90% CI 2-sided [0.1 to 16.7] — Risk difference = (risankizumab - Placebo)
Statistical Analysis 3: Comparison: Substudy 1, Induction Period 1: Double-blind Placebo IV vs Substudy 1, Induction Period 1: Double-blind Risankizumab 1800mg IV; Test type: Superiority; p = 0.0512, Cochran-Mantel-Haenszel — P-value ≤ 0.1; Stratified by baseline corticosteroid use (yes, no) and baseline adapted mayo score (<= 7, > 7); Adjusted Risk Difference = 10.5, 90% CI 2-sided [1.6 to 19.3] — Risk difference = (risankizumab - Placebo)

4. Secondary Outcome: Sub-Study 1: Percentage of Participants Achieving Clinical Remission Per Full Mayo Score in Participants With a Full Mayo Score of 6 to 12 at Baseline
Description: The Mayo score is a tool designed to measure disease activity for ulcerative colitis. The Full Mayo score (FMS) ranges from 0 (normal or inactive disease) to 12 (severe disease) and is calculated as the sum of 4 subscores (stool frequency, rectal bleeding, endoscopy [confirmed by a central reader], and physician's global assessment), each of which ranges from 0 (normal) to 3 (severe disease). Negative changes indicate improvement.
  Clinical remission per FMS is defined as Mayo Score ≤ 2 and no individual subscore > 1.
Time Frame: Week 12
Population: No data was collected.
Arm/Group | Substudy 1, Induction Period 1: Double-blind Placebo IV | Substudy 1, Induction Period 1: Double-blind Risankizumab 600mg IV | Substudy 1, Induction Period 1: Double-blind Risankizumab 1200mg IV | Substudy 1, Induction Period 1: Double-blind Risankizumab 1800mg IV | Substudy 1, Induction Period 1: Open-label Risankizumab 1800mg IV
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Sub-Study 1: Percentage of Participants Achieving Clinical Response Per Adapted Mayo Score
Description: The Adapted Mayo Score is a composite score of UC disease activity based on the following 3 subscores:
  1. Stool frequency subscore (SFS), scored from 0 (normal number of stools) to 3 (5 or more stools more than normal)
  2. Rectal bleeding subscore (RBS), scored from 0 (no blood seen) to 3 (blood alone passed)
  3. Endoscopic subscore, scored from 0 (normal or inactive disease) to 3 (severe disease, spontaneous bleeding, ulceration)
  The overall Adapted Mayo Score ranges from 0 to 9 where higher scores represent more severe disease.
  Clinical response per Adapted Mayo Score was defined as decrease from baseline in Adapted Mayo Score ≥ 2 points and ≥ 30%, plus a decrease in RBS ≥ 1 or an absolute RBS ≤ 1.
Time Frame: Week 12
Population: Includes ITT1A and ITT1B populations.
Measure: Count of Participants; unit: Participants
Arm/Group | Substudy 1, Induction Period 1: Double-blind Placebo IV | Substudy 1, Induction Period 1: Double-blind Risankizumab 600mg IV | Substudy 1, Induction Period 1: Double-blind Risankizumab 1200mg IV | Substudy 1, Induction Period 1: Double-blind Risankizumab 1800mg IV | Substudy 1, Induction Period 1: Open-label Risankizumab 1800mg IV
Number analyzed (Participants) | 60 | 61 | 61 | 58 | 340
Participants | 12 | 26 | 28 | 31 | 157
Statistical Analysis 1: Comparison: Substudy 1, Induction Period 1: Double-blind Placebo IV vs Substudy 1, Induction Period 1: Double-blind Risankizumab 600mg IV; Test type: Superiority; p = 0.0022, Cochran-Mantel-Haenszel — P-value ≤ 0.01; Stratified by baseline corticosteroid use (yes, no) and baseline adapted mayo score (<= 7, > 7); Adjusted Risk Difference = 23.9, 90% CI 2-sided [11.0 to 36.7] — Risk difference = (risankizumab - Placebo)
Statistical Analysis 2: Comparison: Substudy 1, Induction Period 1: Double-blind Placebo IV vs Substudy 1, Induction Period 1: Double-blind Risankizumab 1200mg IV; Test type: Superiority; p = 0.0002, Cochran-Mantel-Haenszel — P-value ≤ 0.001; Stratified by baseline corticosteroid use (yes, no) and baseline adapted mayo score (<= 7, > 7); Adjusted Risk Difference = 28.4, 90% CI 2-sided [15.7 to 41.1] — Risk difference = (risankizumab - Placebo)
Statistical Analysis 3: Comparison: Substudy 1, Induction Period 1: Double-blind Placebo IV vs Substudy 1, Induction Period 1: Double-blind Risankizumab 1800mg IV; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value ≤ 0.001; Stratified by baseline corticosteroid use (yes, no) and baseline adapted mayo score (<= 7, > 7); Adjusted Risk Difference = 33.8, 90% CI 2-sided [20.7 to 46.9] — Risk difference = (risankizumab - Placebo)

6. Secondary Outcome: Sub-Study 1: Percentage of Participants Achieving Clinical Response Per Partial Adapted Mayo Score
Description: Clinical response per Partial Adapted Mayo Score (without endoscopy).
  The Partial Mayo Score is a composite score of UC disease activity based on the following 2 subscores:
  1. Stool frequency subscore (SFS), scored from 0 (normal number of stools) to 3 (5 or more stools more than normal)
  2. Rectal bleeding subscore (RBS), scored from 0 (no blood seen) to 3 (blood alone passed)
  The overall Partial Mayo Score ranges from 0 to 6 with higher scores representing more severe disease.
  Clinical response per Partial Mayo Score is defined as a decrease in Partial Adapted Mayo score >= 1 points and ≥ 30% from Baseline, plus a decrease in RBS ≥ 1 or an absolute RBS ≤ 1.
Time Frame: Week 4
Population: Includes ITT1A and ITT1B populations.
Measure: Count of Participants; unit: Participants
Arm/Group | Substudy 1, Induction Period 1: Double-blind Placebo IV | Substudy 1, Induction Period 1: Double-blind Risankizumab 600mg IV | Substudy 1, Induction Period 1: Double-blind Risankizumab 1200mg IV | Substudy 1, Induction Period 1: Double-blind Risankizumab 1800mg IV | Substudy 1, Induction Period 1: Open-label Risankizumab 1800mg IV
Number analyzed (Participants) | 60 | 61 | 61 | 58 | 340
Participants | 15 | 20 | 28 | 22 | 148
Statistical Analysis 1: Comparison: Substudy 1, Induction Period 1: Double-blind Placebo IV vs Substudy 1, Induction Period 1: Double-blind Risankizumab 600mg IV; Test type: Superiority; p = 0.1842, Cochran-Mantel-Haenszel; Stratified by baseline corticosteroid use (yes, no) and baseline adapted mayo score (<= 7, > 7); Adjusted Risk Difference = 10.2, 90% CI 2-sided [-2.4 to 22.9] — Risk difference = (risankizumab - Placebo)
Statistical Analysis 2: Comparison: Substudy 1, Induction Period 1: Double-blind Placebo IV vs Substudy 1, Induction Period 1: Double-blind Risankizumab 1200mg IV; Test type: Superiority; p = 0.0041, Cochran-Mantel-Haenszel — P-value ≤ 0.01; Stratified by baseline corticosteroid use (yes, no) and baseline adapted mayo score (<= 7, > 7); Adjusted Risk Difference = 23.2, 90% CI 2-sided [9.9 to 36.4] — Risk difference = (risankizumab - Placebo)
Statistical Analysis 3: Comparison: Substudy 1, Induction Period 1: Double-blind Placebo IV vs Substudy 1, Induction Period 1: Double-blind Risankizumab 1800mg IV; Test type: Superiority; p = 0.1117, Cochran-Mantel-Haenszel; Stratified by baseline corticosteroid use (yes, no) and baseline adapted mayo score (<= 7, > 7); Adjusted Risk Difference = 13.1, 90% CI 2-sided [-0.4 to 26.6] — Risk difference = (risankizumab - Placebo)

7. Secondary Outcome: Sub-Study 1: Percentage of Participants Achieving Endoscopic Remission
Description: Endoscopic remission was defined as endoscopy subscore of 0.
Time Frame: Week 12
Population: Includes ITT1A and ITT1B populations.
Measure: Count of Participants; unit: Participants
Arm/Group | Substudy 1, Induction Period 1: Double-blind Placebo IV | Substudy 1, Induction Period 1: Double-blind Risankizumab 600mg IV | Substudy 1, Induction Period 1: Double-blind Risankizumab 1200mg IV | Substudy 1, Induction Period 1: Double-blind Risankizumab 1800mg IV | Substudy 1, Induction Period 1: Open-label Risankizumab 1800mg IV
Number analyzed (Participants) | 60 | 61 | 61 | 58 | 340
Participants | 0 | 5 | 3 | 5 | 22
Statistical Analysis 1: Comparison: Substudy 1, Induction Period 1: Double-blind Placebo IV vs Substudy 1, Induction Period 1: Double-blind Risankizumab 600mg IV; Test type: Superiority; p = 0.0192, Cochran-Mantel-Haenszel — P-value ≤ 0.05; Stratified by baseline corticosteroid use (yes, no) and baseline adapted mayo score (<= 7, > 7); Adjusted Risk Difference = 8.3, 90% CI 2-sided [2.5 to 14.1] — Risk difference = (risankizumab - Placebo)
Statistical Analysis 2: Comparison: Substudy 1, Induction Period 1: Double-blind Placebo IV vs Substudy 1, Induction Period 1: Double-blind Risankizumab 1200mg IV; Test type: Superiority; p = 0.0706, Cochran-Mantel-Haenszel — P-value ≤ 0.1; Stratified by baseline corticosteroid use (yes, no) and baseline adapted mayo score (<= 7, > 7); Adjusted Risk Difference = 4.8, 90% CI 2-sided [0.4 to 9.1] — Risk difference = (risankizumab - Placebo)
Statistical Analysis 3: Comparison: Substudy 1, Induction Period 1: Double-blind Placebo IV vs Substudy 1, Induction Period 1: Double-blind Risankizumab 1800mg IV; Test type: Superiority; p = 0.0170, Cochran-Mantel-Haenszel — P-value ≤ 0.05; Stratified by baseline corticosteroid use (yes, no) and baseline adapted mayo score (<= 7, > 7); Adjusted Risk Difference = 8.7, 90% CI 2-sided [2.7 to 14.6] — Risk difference = (risankizumab - Placebo)

8. Secondary Outcome: Sub-Study 1: Percentage of Participants With Hospitalization
Description: Participants with an event that results in admission to the hospital.
Time Frame: Through Week 12
Population: Includes ITT1A and ITT1B populations.
Measure: Count of Participants; unit: Participants
Arm/Group | Substudy 1, Induction Period 1: Double-blind Placebo IV | Substudy 1, Induction Period 1: Double-blind Risankizumab 600mg IV | Substudy 1, Induction Period 1: Double-blind Risankizumab 1200mg IV | Substudy 1, Induction Period 1: Double-blind Risankizumab 1800mg IV | Substudy 1, Induction Period 1: Open-label Risankizumab 1800mg IV
Number analyzed (Participants) | 60 | 61 | 61 | 58 | 340
Participants | 5 | 6 | 4 | 3 | 19
Statistical Analysis 1: Comparison: Substudy 1, Induction Period 1: Double-blind Placebo IV vs Substudy 1, Induction Period 1: Double-blind Risankizumab 600mg IV; Test type: Superiority; p = 0.7737, Chi-squared; P value for comparisons between treatment groups and placebo group using chi-square test or Fisher's exact test
Statistical Analysis 2: Comparison: Substudy 1, Induction Period 1: Double-blind Placebo IV vs Substudy 1, Induction Period 1: Double-blind Risankizumab 1200mg IV; Test type: Superiority; p = 0.7432, Fisher Exact; P value for comparisons between treatment groups and placebo group using chi-square test or Fisher's exact test
Statistical Analysis 3: Comparison: Substudy 1, Induction Period 1: Double-blind Placebo IV vs Substudy 1, Induction Period 1: Double-blind Risankizumab 1800mg IV; Test type: Superiority; p = 0.7172, Fisher Exact; P value for comparisons between treatment groups and placebo group using chi-square test or Fisher's exact test

9. Secondary Outcome: Sub-Study 1: Percentage of Participants Achieving Histologic Endoscopic Mucosal Remission (HEMR)
Description: Mucosal healing defined as endoscopic and histologic remission.
  Mucosal healing is defined as an endoscopic score of 0 and Geboes score < 2.0. The endoscopic subscore ranges from 0 (normal or inactive disease) to 3 (severe disease with spontaneous bleeding, ulceration).
  The Geboes histologic index includes seven histological features (architectural change, chronic inflammatory infiltrate, lamina propria neutrophils and eosinophils, neutrophils in epithelium, crypt destruction and erosion or ulcers). The Geboes score has 6 grades, each with 3-5 subgrades: Grade 0, structural change only; Grade 1, chronic inflammation; Grade 2, lamina propria neutrophils and eosinophils; Grade 3, neutrophils in epithelium; Grade 4, crypt destruction; and Grade 5, erosions or ulceration.
Time Frame: Week 12
Population: Includes ITT1A and ITT1B populations.
Measure: Count of Participants; unit: Participants
Arm/Group | Substudy 1, Induction Period 1: Double-blind Placebo IV | Substudy 1, Induction Period 1: Double-blind Risankizumab 600mg IV | Substudy 1, Induction Period 1: Double-blind Risankizumab 1200mg IV | Substudy 1, Induction Period 1: Double-blind Risankizumab 1800mg IV | Substudy 1, Induction Period 1: Open-label Risankizumab 1800mg IV
Number analyzed (Participants) | 60 | 61 | 61 | 58 | 340
Participants | 0 | 3 | 2 | 1 | 10
Statistical Analysis 1: Comparison: Substudy 1, Induction Period 1: Double-blind Placebo IV vs Substudy 1, Induction Period 1: Double-blind Risankizumab 600mg IV; Test type: Superiority; p = 0.0722, Cochran-Mantel-Haenszel — P-value ≤ 0.1; Stratified by baseline corticosteroid use (yes, no) and baseline adapted mayo score (<= 7, > 7); Adjusted Risk Difference = 4.7, 90% CI 2-sided [0.4 to 9.0] — Risk difference = (risankizumab - Placebo)
Statistical Analysis 2: Comparison: Substudy 1, Induction Period 1: Double-blind Placebo IV vs Substudy 1, Induction Period 1: Double-blind Risankizumab 1200mg IV; Test type: Superiority; p = 0.1480, Cochran-Mantel-Haenszel; Stratified by baseline corticosteroid use (yes, no) and baseline adapted mayo score (<= 7, > 7); Adjusted Risk Difference = 3.1, 90% CI 2-sided [-0.4 to 6.6] — Risk difference = (risankizumab - Placebo)
Statistical Analysis 3: Comparison: Substudy 1, Induction Period 1: Double-blind Placebo IV vs Substudy 1, Induction Period 1: Double-blind Risankizumab 1800mg IV; Test type: Superiority; p = 0.3042, Cochran-Mantel-Haenszel; Stratified by baseline corticosteroid use (yes, no) and baseline adapted mayo score (<= 7, > 7); Adjusted Risk Difference = 1.7, 90% CI 2-sided [-1.0 to 4.5] — Risk difference = (risankizumab - Placebo)

10. Secondary Outcome: Sub-Study 1: Change in Ulcerative Colitis Symptom Questionnaire (UC-SQ)
Description: The US-SQ is a patient questionnaire to assess severity of Ulcerative Colitis (UC) related gastrointestinal symptoms (e.g., frequent bowel movements, abdominal pain, cramping) and non-gastrointestinal symptoms (e.g., joint pain and sleep difficulties).
  It consists of 17 questions and each question is answered on a scale from can be answered on a scale from 1 (Not at all/ never) to 5 (Very much/Always) with overall symptom score range from 17 to 85. A lower score indicates lower UC severity.
Time Frame: Baseline Through Week 12
Population: Includes ITT1A and ITT1B participants with data available for analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Substudy 1, Induction Period 1: Double-blind Placebo IV | Substudy 1, Induction Period 1: Double-blind Risankizumab 600mg IV | Substudy 1, Induction Period 1: Double-blind Risankizumab 1200mg IV | Substudy 1, Induction Period 1: Double-blind Risankizumab 1800mg IV | Substudy 1, Induction Period 1: Open-label Risankizumab 1800mg IV
Number analyzed (Participants) | 50 | 52 | 56 | 53 | 286
units on a scale | -7.4 (1.53) | -13.8 (1.50) | -15.6 (1.46) | -15.1 (1.51) | -17.1 (0.58)
Statistical Analysis 1: Comparison: Substudy 1, Induction Period 1: Double-blind Placebo IV vs Substudy 1, Induction Period 1: Double-blind Risankizumab 600mg IV; Test type: Superiority; p = 0.0030, Mixed-effect model repeated measurement — P-value ≤ 0.01; Least Squares (LS) Mean Difference = -6.4, 90% CI 2-sided [-9.94 to -2.89], Standard Error of Mean 2.13
Statistical Analysis 2: Comparison: Substudy 1, Induction Period 1: Double-blind Placebo IV vs Substudy 1, Induction Period 1: Double-blind Risankizumab 1200mg IV; Test type: Superiority; p = 0.0001, Mixed-effect model repeated measurement — P-value ≤ 0.001; Least Squares (LS) Mean Difference = -8.2, 90% CI 2-sided [-11.67 to -4.71], Standard Error of Mean 2.11
Statistical Analysis 3: Comparison: Substudy 1, Induction Period 1: Double-blind Placebo IV vs Substudy 1, Induction Period 1: Double-blind Risankizumab 1800mg IV; Test type: Superiority; p = 0.0004, Mixed-effect model repeated measurement — P-value ≤ 0.001; Least Squares (LS) Mean Difference = -7.7, 90% CI 2-sided [-11.27 to -4.19], Standard Error of Mean 2.14

11. Secondary Outcome: Sub-Study 1: Change in Inflammatory Bowel Disease Questionnaire (IBDQ)
Description: The IBDQ is used to assess the quality of life of patients with inflammatory bowel disease.
  The IBDQ is a 32-item (ranges 1 - 7) self-report questionnaire for patients with IBD to evaluate the patient reported outcomes across 4 dimensions: bowel symptoms (loose stools, abdominal pain), systemic symptoms (fatigue, altered sleep pattern), social function (work attendance, need to cancel social events), and emotional function (anger, depression, irritability).
  The IBDQ total Score ranges from 32 to 224 with a higher score indicating better outcome.
Time Frame: Baseline Through Week 12
Population: Includes ITT1A and ITT1B participants with data available for analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Substudy 1, Induction Period 1: Double-blind Placebo IV | Substudy 1, Induction Period 1: Double-blind Risankizumab 600mg IV | Substudy 1, Induction Period 1: Double-blind Risankizumab 1200mg IV | Substudy 1, Induction Period 1: Double-blind Risankizumab 1800mg IV | Substudy 1, Induction Period 1: Open-label Risankizumab 1800mg IV
Number analyzed (Participants) | 51 | 55 | 59 | 54 | 305
units on a scale | 20.1 (4.67) | 37.4 (4.56) | 40.3 (4.38) | 40.0 (4.55) | 49.5 (1.86)
Statistical Analysis 1: Comparison: Substudy 1, Induction Period 1: Double-blind Placebo IV vs Substudy 1, Induction Period 1: Double-blind Risankizumab 600mg IV; Test type: Superiority; p = 0.0081, Mixed-effect model repeated measurement — P-value ≤ 0.01; Least Squares (LS) Mean Difference = 17.3, 90% CI 2-sided [6.61 to 28], Standard Error of Mean 6.47
Statistical Analysis 2: Comparison: Substudy 1, Induction Period 1: Double-blind Placebo IV vs Substudy 1, Induction Period 1: Double-blind Risankizumab 1200mg IV; Test type: Superiority; p = 0.0017, Mixed-effect model repeated measurement — P-value ≤ 0.01; Least Squares (LS) Mean Difference = 20.3, 90% CI 2-sided [9.74 to 30.79], Standard Error of Mean 6.37
Statistical Analysis 3: Comparison: Substudy 1, Induction Period 1: Double-blind Placebo IV vs Substudy 1, Induction Period 1: Double-blind Risankizumab 1800mg IV; Test type: Superiority; p = 0.0024, Mixed-effect model repeated measurement — P-value ≤ 0.01; Least Squares (LS) Mean Difference = 19.9, 90% CI 2-sided [9.22 to 30.67], Standard Error of Mean 6.49

12. Secondary Outcome: Sub-Study 1: Change From Baseline in Short Form-36 (SF-36) - Physical Component
Description: The SF-36 (Version 2) is a self-administered, health-related survey that measures the impact of disease on overall quality of life during the past 4 weeks. SF-36 consists of 36 questions covering 8 health domains: physical functioning, bodily pain, role limitations due to physical problems and emotional problems, general health, mental health, social functioning, vitality, and 2 component scores (mental [MCS] and physical [PCS]). MCS consisted of social functioning, vitality, mental health, and role-emotional scales. PCS consisted of physical functioning, bodily pain, role-physical, and general health scales. Each domain is scored by summing the individual items and transforming the scores into a 0 (poorest health) to 100 (best health) scale with higher scores indicating better health status or functioning.
Time Frame: Baseline Through Week 12
Population: Includes ITT1A and ITT1B participants with data available for analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Substudy 1, Induction Period 1: Double-blind Placebo IV | Substudy 1, Induction Period 1: Double-blind Risankizumab 600mg IV | Substudy 1, Induction Period 1: Double-blind Risankizumab 1200mg IV | Substudy 1, Induction Period 1: Double-blind Risankizumab 1800mg IV | Substudy 1, Induction Period 1: Open-label Risankizumab 1800mg IV
Number analyzed (Participants) | 51 | 54 | 59 | 54 | 298
units on a scale | 3.904 (0.8907) | 5.112 (0.8751) | 6.350 (0.8341) | 6.296 (0.8675) | 7.719 (0.3929)
Statistical Analysis 1: Comparison: Substudy 1, Induction Period 1: Double-blind Placebo IV vs Substudy 1, Induction Period 1: Double-blind Risankizumab 600mg IV; Test type: Superiority; p = 0.3315, Mixed-effect model repeated measurement; Least Squares (LS) Mean Difference = 1.208, 90% CI 2-sided [-0.8429 to 3.2596]
Statistical Analysis 2: Comparison: Substudy 1, Induction Period 1: Double-blind Placebo IV vs Substudy 1, Induction Period 1: Double-blind Risankizumab 1200mg IV; Test type: Superiority; p = 0.0451, Mixed-effect model repeated measurement — P-value ≤ 0.05; LS Mean of Difference = 2.447, 90% CI 2-sided [0.4415 to 4.4519]
Statistical Analysis 3: Comparison: Substudy 1, Induction Period 1: Double-blind Placebo IV vs Substudy 1, Induction Period 1: Double-blind Risankizumab 1800mg IV; Test type: Superiority; p = 0.0543, Mixed-effect model repeated measurement — P-value ≤ 0.1; LS Mean of Difference = 2.392, 90% CI 2-sided [0.3498 to 4.4352]

13. Secondary Outcome: Sub-Study 1: Change From Baseline in Short Form-36 (SF-36) - Mental Component
Description: as for outcome 12
Time Frame: Baseline through Week 12
Population: Includes ITT1A and ITT1B participants with data available for analysis.
Measure: Least Squares Mean (Standard Error); unit: unites on a scale
Arm/Group | Substudy 1, Induction Period 1: Double-blind Placebo IV | Substudy 1, Induction Period 1: Double-blind Risankizumab 600mg IV | Substudy 1, Induction Period 1: Double-blind Risankizumab 1200mg IV | Substudy 1, Induction Period 1: Double-blind Risankizumab 1800mg IV | Substudy 1, Induction Period 1: Open-label Risankizumab 1800mg IV
Number analyzed (Participants) | 51 | 54 | 59 | 54 | 298
unites on a scale | 3.094 (1.2533) | 6.756 (1.2319) | 7.284 (1.1739) | 5.442 (1.2185) | 7.777 (0.4777)
Statistical Analysis 1: Comparison: Substudy 1, Induction Period 1: Double-blind Placebo IV vs Substudy 1, Induction Period 1: Double-blind Risankizumab 600mg IV; Test type: Superiority; p = 0.0367, Mixed-effect model repeated measurement — P-value <= 0.1; LS Mean of Difference = 3.662, 90% CI 2-sided [0.7841 to 6.5402] — P-value for test of difference between each Risankizumab dose group and placebo for mean change from baseline using the mixed-effect repeated measure model The unstructured covariance structure was used to estimate within subject errors
Statistical Analysis 2: Comparison: Substudy 1, Induction Period 1: Double-blind Placebo IV vs Substudy 1, Induction Period 1: Double-blind Risankizumab 1200mg IV; Test type: Superiority; p = 0.0151, Mixed-effect model repeated measurement — P-value <= 0.05; LS Mean of Difference = 4.190, 90% CI 2-sided [1.3656 to 7.0144] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 3: Comparison: Substudy 1, Induction Period 1: Double-blind Placebo IV vs Substudy 1, Induction Period 1: Double-blind Risankizumab 1800mg IV; Test type: Superiority; p = 0.1795, Mixed-effect model repeated measurement; LS Mean of Difference = 2.348, 90% CI 2-sided [-0.5322 to 5.2281] — [estimate comment as in outcome 13, analysis 1]

14. Secondary Outcome: Sub-Study 1: Change in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue)
Description: The FACIT-Fatigue Scale is a validated self-administered 13-item tool that measures an individual's level of fatigue during their usual daily activities over the past 7 days. Each of the fatigue and impact of fatigue items are measured on a four-point Likert scale.
  0 = not at all
  1. = a little bit
  2. = somewhat
  3. = quite a bit
  4. = very much
  The FACIT Fatigue Scale is the sum of the individual 13 scores and ranges from 0 to 52 where higher scores indicate better the quality of life. A positive change from baseline indicates improvement.
Time Frame: Baseline Through Week 12
Population: Includes ITT1A and ITT1B participants with data available for analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Substudy 1, Induction Period 1: Double-blind Placebo IV | Substudy 1, Induction Period 1: Double-blind Risankizumab 600mg IV | Substudy 1, Induction Period 1: Double-blind Risankizumab 1200mg IV | Substudy 1, Induction Period 1: Double-blind Risankizumab 1800mg IV | Substudy 1, Induction Period 1: Open-label Risankizumab 1800mg IV
Number analyzed (Participants) | 51 | 54 | 59 | 54 | 298
units on a scale | 3.7 (1.37) | 7.6 (1.35) | 9.0 (1.29) | 8.3 (1.33) | 10.7 (0.54)
Statistical Analysis 1: Comparison: Substudy 1, Induction Period 1: Double-blind Placebo IV vs Substudy 1, Induction Period 1: Double-blind Risankizumab 600mg IV; Test type: Superiority; p = 0.0422, Mixed-effect model repeated measurement — P-value ≤ 0.05; Least Squares (LS) Mean Difference = 3.9, 90% CI 2-sided [0.75 to 7.06], Standard Error of Mean 1.91
Statistical Analysis 2: Comparison: Substudy 1, Induction Period 1: Double-blind Placebo IV vs Substudy 1, Induction Period 1: Double-blind Risankizumab 1200mg IV; Test type: Superiority; p = 0.0049, Mixed-effect model repeated measurement — P-value ≤ 0.01; Least Squares (LS) Mean Difference = 5.3, 90% CI 2-sided [2.23 to 8.42], Standard Error of Mean 1.87
Statistical Analysis 3: Comparison: Substudy 1, Induction Period 1: Double-blind Placebo IV vs Substudy 1, Induction Period 1: Double-blind Risankizumab 1800mg IV; Test type: Superiority; p = 0.0156, Mixed-effect model repeated measurement — P-value ≤ 0.05; Least Squares (LS) Mean Difference = 4.6, 90% CI 2-sided [1.50 to 7.80], Standard Error of Mean 1.91

15. Secondary Outcome: Sub-Study 1: Percentage of Participants Undergoing Ulcerative Colitis (UC)-Related Surgeries
Description: Participants who underwent surgery related to UC.
Time Frame: Through Week 12
Population: Includes ITT1A and ITT1B populations.
Measure: Count of Participants; unit: Participants
Arm/Group | Substudy 1, Induction Period 1: Double-blind Placebo IV | Substudy 1, Induction Period 1: Double-blind Risankizumab 600mg IV | Substudy 1, Induction Period 1: Double-blind Risankizumab 1200mg IV | Substudy 1, Induction Period 1: Double-blind Risankizumab 1800mg IV | Substudy 1, Induction Period 1: Open-label Risankizumab 1800mg IV
Number analyzed (Participants) | 60 | 61 | 61 | 58 | 340
Participants | 0 | 1 | 0 | 0 | 7
Statistical Analysis 1: Comparison: Substudy 1, Induction Period 1: Double-blind Placebo IV vs Substudy 1, Induction Period 1: Double-blind Risankizumab 600mg IV; Note: ITT1A includes all randomized subjects who received at least one dose of study drug during Induction Period 1 from Sub-Study 1; Test type: Superiority; p = 1, Fisher Exact — P-Value for comparisons between treatment groups and placebo group using Fisher's exact test

16. Secondary Outcome: Sub-Study 2: Percentage of Participants Achieving Clinical Response Per Adapted Mayo Score
Description: The Adapted Mayo Score is a composite score of UC disease activity based on the following 3 subscores:
  1. Stool frequency subscore (SFS), scored from 0 (normal number of stools) to 3 (5 or more stools more than normal)
  2. Rectal bleeding subscore (RBS), scored from 0 (no blood seen) to 3 (blood alone passed)
  3. Endoscopic subscore, scored from 0 (normal or inactive disease) to 3 (severe disease, spontaneous bleeding, ulceration)
  The overall Adapted Mayo Score ranges from 0 to 9 where higher scores represent more severe disease.
  Clinical Response is defined as a decrease from baseline in the Adapted Mayo Score ≥ 2 points and ≥ 30% from baseline, and a decrease in RBS ≥ 1 or an absolute RBS ≤ 1).
Time Frame: Week 12
Population: ITT2 includes all randomized subjects who received at least one dose of study drug during Induction Period 1 from Sub-Study 2.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Substudy 2, Induction Period 1: Double-blind Placebo IV | Substudy 2, Induction Period 1: Double-blind Risankizumab 1200mg IV
Number analyzed (Participants) | 325 | 650
percentage of participants | 35.7 [30.5 to 40.9] | 64.3 [60.6 to 67.9]
Statistical Analysis 1: Comparison: Substudy 2, Induction Period 1: Double-blind Placebo IV vs Substudy 2, Induction Period 1: Double-blind Risankizumab 1200mg IV; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Statistical significance is determined via the graphical multiple testing procedure controlling the overall type I error rate of primary and key secondary endpoints at the 0.05 level; Adjusted Risk Difference = 28.6, 95% CI 2-sided [22.3 to 34.8] — Between-group diff. and 95% CI calculated using Mantel-Haenszel common rate difference

17. Secondary Outcome: Sub-Study 2: Percentage of Participants Achieving Endoscopic Improvement
Description: Endoscopic Improvement is defined as an endoscopic subscore of 0 or 1.
  Endoscopies were assessed by a blinded central reader and scored according to the following scale: 0 = Normal or inactive disease; 1 = Mild disease (erythema, decreased vascular pattern); 2 = Moderate disease (marked erythema, lack of vascular pattern, any friability, erosions); 3 = Severe disease (spontaneous bleeding, ulceration).
Time Frame: Week 12
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Substudy 2, Induction Period 1: Double-blind Placebo IV | Substudy 2, Induction Period 1: Double-blind Risankizumab 1200mg IV
Number analyzed (Participants) | 325 | 650
percentage of participants | 12.1 [8.5 to 15.6] | 36.5 [32.8 to 40.2]
Statistical Analysis 1: Comparison: Substudy 2, Induction Period 1: Double-blind Placebo IV vs Substudy 2, Induction Period 1: Double-blind Risankizumab 1200mg IV; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]; Adjusted Risk Difference = 24.3, 95% CI 2-sided [19.3 to 29.4] — Between-group diff. and 95% CI calculated using Mantel-Haenszel common rate difference. (Greenland and Robins (1985))

18. Secondary Outcome: Sub-Study 2: Percentage of Participants Achieving Histologic Endoscopic Mucosal Improvement (HEMI)
Description: Histologic-Endoscopic Mucosal Improvement is defined as an endoscopic subscore of 0 or 1 without evidence of friability and a Geboes score ≤ 3.1.
  The endoscopic subscore ranges from 0 (normal or inactive disease) to 3 (severe disease with spontaneous bleeding, ulceration).
  The Geboes histologic index includes seven histological features (architectural change, chronic inflammatory infiltrate, lamina propria neutrophils and eosinophils, neutrophils in epithelium, crypt destruction and erosion or ulcers).
  The Geboes score has 6 grades, each with 3-5 subgrades: Grade 0, structural change only; Grade 1, chronic inflammation; Grade 2, lamina propria neutrophils and eosinophils; Grade 3, neutrophils in epithelium; Grade 4, crypt destruction; and Grade 5, erosions or ulceration.
Time Frame: Week 12
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Substudy 2, Induction Period 1: Double-blind Placebo IV | Substudy 2, Induction Period 1: Double-blind Risankizumab 1200mg IV
Number analyzed (Participants) | 325 | 650
percentage of participants | 7.7 [4.8 to 10.6] | 24.5 [21.2 to 27.8]
Statistical Analysis 1: Comparison: Substudy 2, Induction Period 1: Double-blind Placebo IV vs Substudy 2, Induction Period 1: Double-blind Risankizumab 1200mg IV; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]; Adjusted Risk Difference = 16.6, 95% CI 2-sided [12.3 to 21.0] — Between-group diff. and 95% CI calculated using Mantel-Haenszel common rate difference. (Greenland and Robins (1985))

19. Secondary Outcome: Sub-Study 2: Percentage of Participants Achieving Endoscopic Remission
Description: Endoscopic remission per endoscopy subscore.
  Endoscopic Remission: endoscopic subscore = 0.
Time Frame: Week 12
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Substudy 2, Induction Period 1: Double-blind Placebo IV | Substudy 2, Induction Period 1: Double-blind Risankizumab 1200mg IV
Number analyzed (Participants) | 325 | 650
percentage of participants | 3.4 [1.4 to 5.4] | 10.6 [8.2 to 13.0]
Statistical Analysis 1: Comparison: Substudy 2, Induction Period 1: Double-blind Placebo IV vs Substudy 2, Induction Period 1: Double-blind Risankizumab 1200mg IV; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]; Adjusted Risk Difference = 7.2, 95% CI 2-sided [4.2 to 10.2] — Between-group diff. and 95% CI calculated using Mantel-Haenszel common rate difference. (Greenland and Robins (1985))

20. Secondary Outcome: Sub-Study 2: Percentage of Participants Achieving Clinical Response Per Partial Adapted Mayo Score at Week 4
Description: Clinical response per Partial Adapted Mayo Score (without endoscopy).
  The Partial Mayo Score is a composite score of UC disease activity based on the following 2 subscores:
  1. Stool frequency subscore (SFS), scored from 0 (normal number of stools) to 3 (5 or more stools more than normal)
  2. Rectal bleeding subscore (RBS), scored from 0 (no blood seen) to 3 (blood alone passed)
  The overall Partial Mayo Score ranges from 0 to 6 with higher scores representing more severe disease.
  Clinical Response per Partial Mayo Score is defined as a decrease in Partial Adapted Mayo Score ≥ 1 points and ≥ 30% from Baseline, plus a decrease in RBS ≥ 1 or an absolute RBS ≤ 1.
Time Frame: Week 4
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Substudy 2, Induction Period 1: Double-blind Placebo IV | Substudy 2, Induction Period 1: Double-blind Risankizumab 1200mg IV
Number analyzed (Participants) | 325 | 650
percentage of participants | 30.5 [25.5 to 35.5] | 52.2 [48.3 to 56.0]
Statistical Analysis 1: Comparison: Substudy 2, Induction Period 1: Double-blind Placebo IV vs Substudy 2, Induction Period 1: Double-blind Risankizumab 1200mg IV; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]; Adjusted Risk Difference = 21.8, 95% CI 2-sided [15.6 to 28.1] — Between-group diff. and 95% CI calculated using Mantel-Haenszel common rate difference. (Greenland and Robins (1985))

21. Secondary Outcome: Sub-Study 2: Percentage of Participants Achieving No Bowel Urgency
Description: Percentage of participants who reported no bowel urgency. Bowel urgency was assessed by participants in a subject diary completed once a day.
Time Frame: Week 12
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Substudy 2, Induction Period 1: Double-blind Placebo IV | Substudy 2, Induction Period 1: Double-blind Risankizumab 1200mg IV
Number analyzed (Participants) | 325 | 650
percentage of participants | 27.7 [22.8 to 32.6] | 44.1 [40.3 to 47.9]
Statistical Analysis 1: Comparison: Substudy 2, Induction Period 1: Double-blind Placebo IV vs Substudy 2, Induction Period 1: Double-blind Risankizumab 1200mg IV; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]; Adjusted Risk Difference = 16.3, 95% CI 2-sided [10.3 to 22.4] — Between-group diff. and 95% CI calculated using Mantel-Haenszel common rate difference. (Greenland and Robins (1985))

22. Secondary Outcome: Sub-Study 2: Percentage of Participants Achieving No Abdominal Pain
Description: Percentage of participants who reported no abdominal pain. Abdominal pain was assessed by participants in a subject diary completed once a day.
Time Frame: Week 12
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Substudy 2, Induction Period 1: Double-blind Placebo IV | Substudy 2, Induction Period 1: Double-blind Risankizumab 1200mg IV
Number analyzed (Participants) | 325 | 650
percentage of participants | 26.5 [21.7 to 31.3] | 35.8 [32.1 to 39.4]
Statistical Analysis 1: Comparison: Substudy 2, Induction Period 1: Double-blind Placebo IV vs Substudy 2, Induction Period 1: Double-blind Risankizumab 1200mg IV; Test type: Superiority; p = 0.0021, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]; Adjusted Risk Difference = 9.3, 95% CI 2-sided [3.4 to 15.3] — Between-group diff. and 95% CI calculated using Mantel-Haenszel common rate difference. (Greenland and Robins (1985))

23. Secondary Outcome: Sub-Study 2: Percentage of Participants Achieving Histologic Endoscopic Mucosal Remission (HEMR): Endoscopy Subscore of 0 and Geboes Score < 2.0) at Week 12
Description: as for outcome 9
Time Frame: Week 12
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Substudy 2, Induction Period 1: Double-blind Placebo IV | Substudy 2, Induction Period 1: Double-blind Risankizumab 1200mg IV
Number analyzed (Participants) | 325 | 650
percentage of participants | 0.6 [0.0 to 1.5] | 6.3 [4.4 to 8.2]
Statistical Analysis 1: Comparison: Substudy 2, Induction Period 1: Double-blind Placebo IV vs Substudy 2, Induction Period 1: Double-blind Risankizumab 1200mg IV; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]; Adjusted Risk Difference = 5.6, 95% CI 2-sided [3.5 to 7.7] — Between-group diff. and 95% CI calculated using Mantel-Haenszel common rate difference. (Greenland and Robins (1985))

24. Secondary Outcome: Sub-Study 2: Change in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue)
Description: as for outcome 14
Time Frame: Baseline to Week 12
Population: Includes ITT2 participants with data available for analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Substudy 2, Induction Period 1: Double-blind Placebo IV | Substudy 2, Induction Period 1: Double-blind Risankizumab 1200mg IV
Number analyzed (Participants) | 308 | 614
units on a scale | 3.3 [2.12 to 4.50] | 7.9 [7.03 to 8.69]
Statistical Analysis 1: Comparison: Substudy 2, Induction Period 1: Double-blind Placebo IV vs Substudy 2, Induction Period 1: Double-blind Risankizumab 1200mg IV; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 16, analysis 1]; Least Squares (LS) Mean Difference = 4.5, 95% CI 2-sided [3.13 to 5.97] — Between-group diff. and 95% CI calculated using ANCOVA/MMRM with RTB-MI for continuous endpoints

25. Secondary Outcome: Sub-Study 2: Change in Inflammatory Bowel Disease Questionnaire (IBDQ) Total Score
Description: as for outcome 11
Time Frame: Baseline to Week 12
Population: Includes ITT2 participants with data available for analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Substudy 2, Induction Period 1: Double-blind Placebo IV | Substudy 2, Induction Period 1: Double-blind Risankizumab 1200mg IV
Number analyzed (Participants) | 310 | 619
units on a scale | 24.3 [20.19 to 28.46] | 42.6 [39.72 to 45.57]
Statistical Analysis 1: Comparison: Substudy 2, Induction Period 1: Double-blind Placebo IV vs Substudy 2, Induction Period 1: Double-blind Risankizumab 1200mg IV; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 16, analysis 1]; Least Squares (LS) Mean Difference = 18.3, 95% CI 2-sided [13.38 to 23.25] — Between-group diff. and 95% CI calculated using ANCOVA/MMRM with RTB-MI for continuous endpoints

26. Secondary Outcome: Sub-Study 2: Occurrence of UC-related Hospitalizations
Description: Participants with an UC-related event that results in admission to the hospital.
Time Frame: Baseline Through Week 12
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Substudy 2, Induction Period 1: Double-blind Placebo IV | Substudy 2, Induction Period 1: Double-blind Risankizumab 1200mg IV
Number analyzed (Participants) | 325 | 650
percentage of participants | 5.5 [3.1 to 8.0] | 0.8 [0.1 to 1.4]
Statistical Analysis 1: Comparison: Substudy 2, Induction Period 1: Double-blind Placebo IV vs Substudy 2, Induction Period 1: Double-blind Risankizumab 1200mg IV; Test type: Superiority; p < 0.0001, Chi-squared — [p-value comment as in outcome 16, analysis 1]; Risk Difference (RD) = -4.8, 95% CI 2-sided [-7.3 to -2.2] — 95% CI for treatment differences is based on normal approximation of the binomial proportions

27. Secondary Outcome: Sub-Study 2: Percentage of Participants Achieving No Nocturnal Bowel Movements
Description: Percentage of participants who reported no nocturnal bowel movements.
Time Frame: Week 12
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Substudy 2, Induction Period 1: Double-blind Placebo IV | Substudy 2, Induction Period 1: Double-blind Risankizumab 1200mg IV
Number analyzed (Participants) | 325 | 650
percentage of participants | 43.1 [37.7 to 48.5] | 67.3 [63.7 to 70.9]
Statistical Analysis 1: Comparison: Substudy 2, Induction Period 1: Double-blind Placebo IV vs Substudy 2, Induction Period 1: Double-blind Risankizumab 1200mg IV; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]; Adjusted Risk Difference = 24.2, 95% CI 2-sided [17.9 to 30.5] — Between-group diff. and 95% CI calculated using Mantel-Haenszel common rate difference. (Greenland and Robins (1985))

28. Secondary Outcome: Sub-Study 2: Percentage of Participants Achieving No Tenesmus
Description: Percentage of participants who reported no tenesmus.
Time Frame: Week 12
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Substudy 2, Induction Period 1: Double-blind Placebo IV | Substudy 2, Induction Period 1: Double-blind Risankizumab 1200mg IV
Number analyzed (Participants) | 325 | 650
percentage of participants | 30.2 [25.2 to 35.1] | 48.7 [44.9 to 52.6]
Statistical Analysis 1: Comparison: Substudy 2, Induction Period 1: Double-blind Placebo IV vs Substudy 2, Induction Period 1: Double-blind Risankizumab 1200mg IV; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]; Adjusted Risk Difference = 18.6, 95% CI 2-sided [12.4 to 24.8] — Between-group diff. and 95% CI calculated using Mantel-Haenszel common rate difference

29. Secondary Outcome: Sub-Study 2: Change in Number of Fecal Incontinence Episodes Per Week
Description: Change in number of fecal incontinence episodes per week.
Time Frame: Baseline to Week 12
Population: Includes ITT2 participants with data available for analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: Fecal Incontinence Episodes/ week
Arm/Group | Substudy 2, Induction Period 1: Double-blind Placebo IV | Substudy 2, Induction Period 1: Double-blind Risankizumab 1200mg IV
Number analyzed (Participants) | 288 | 602
Fecal Incontinence Episodes/ week | -2.213 [-2.8526 to -1.5726] | -3.839 [-4.2687 to -3.4099]
Statistical Analysis 1: Comparison: Substudy 2, Induction Period 1: Double-blind Placebo IV vs Substudy 2, Induction Period 1: Double-blind Risankizumab 1200mg IV; Test type: Superiority; p < 0.0001, Mixed-Effect Model Repeated Measures — [p-value comment as in outcome 16, analysis 1]; Least Squares (LS) Mean Difference = -1.627, 95% CI 2-sided [-2.3846 to -0.8689] — Between-group diff. and 95% CI calculated using ANCOVA/MMRM with RTB-MI for continuous endpoints

30. Secondary Outcome: Sub-Study 2: Change in Number of Days Per Week With Sleep Interrupted Due to UC Symptoms
Description: Change from baseline in number of days per week with sleep interrupted due to UC symptoms.
Time Frame: Baseline to Week 12
Population: Includes ITT2 participants with data available for analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: days
Arm/Group | Substudy 2, Induction Period 1: Double-blind Placebo IV | Substudy 2, Induction Period 1: Double-blind Risankizumab 1200mg IV
Number analyzed (Participants) | 288 | 602
days | -1.505 [-1.7969 to -1.2122] | -2.485 [-2.6872 to -2.2831]
Statistical Analysis 1: Comparison: Substudy 2, Induction Period 1: Double-blind Placebo IV vs Substudy 2, Induction Period 1: Double-blind Risankizumab 1200mg IV; Test type: Superiority; p < 0.0001, Mixed-Effect Model Repeated Measures — [p-value comment as in outcome 16, analysis 1]; Least Squares (LS) Mean Difference = -0.981, 95% CI 2-sided [-1.3285 to -0.6326] — Between-group diff. and 95% CI calculated using ANCOVA/MMRM with RTB-MI for continuous endpoints

ADVERSE EVENTS:
Time Frame: In S1P1, median time on follow-up was 86, 86, 85, 87, & 87 days(d) for S1P1 DB-PboIV, S1P1 DB-Risankizumab(Risa) 600mgIV, S1P1 DB-Risa 1200mgIV, S1P1 DB-Risa 1800mgIV, and S1P1 OL-Risa 1800mgIV; respectively. In S1P2, median time on follow-up was 87, 106, 93 and 93 d for arms S1P2 DB -Risa 1800mgIVPbo, S1P2 DB-Risa1800mgIV, S1P2 DB-Risa 180mgSC, and S1P2 DB-Risa 360mgSC; respectively. In S2P1, median time on follow-up was 87 and 89d for arms S2P1 DB-PboIV, S2P1 DB Risa1200mgIV, respectively.
Description: In S2P2, median time on follow-up was 143.5, 159, 197and 193d for arms, S2P2 DB-Risa1200mgIVPbo, S2P2 DB-Risa 1200mgIV, S2P2 DB-Risa 180mgSC, and S2P2 DB-Risa 360mgSC; respectively. Safety Events were categorized according to arm subjects were dosed; N=3; 1 subject dosed differently in period S1P1. This subject was assigned into Risa 1800mg IV PbO group in S1P2 (Participant Flow) based on randomization in S1P1, but classified into Risa 1800mg IV S1P2 based on the treatment received in S1P1.
Groups:
- Substudy 1, Induction Period 1: Double-blind Placebo IV: Participants randomized to receive placebo for risankizumab administered by intravenous (IV) infusion.
  1 participant assigned to Placebo IV was dosed with Risankizumab 600 mg IV and is counted in that arm.
- Substudy 1, Induction Period 1: Double-blind Risankizumab 600mg IV: Participants randomized to receive risankizumab 600mg administered by intravenous (IV) infusion.
  1 participant assigned to Placebo IV was dosed with Risankizumab 600 mg IV and is counted in this arm.
- Substudy 1, Induction Period 1: Openlabel Risankizumab 1800mg IV: Participants receive risankizumab 1800mg administered by intravenous (IV) infusion.
- Substudy 1, Induction Period 2: Double-blind Risankizumab 1800mg IV Pbo: Participants who received placebo with inadequate response in Induction 1 receive risankizumab 1800mg administered by intravenous (IV) infusion in Induction 2.
  1 subject was dosed differently in period S1P1 (assigned to Pbo IV but dosed with Risa 600mg IV). This subject was classified into Risa 1800mg IV vs IV PbO based on the treatment received in S1P1.
- Substudy 1, Induction Period 2: Double-blind Risankizumab 1800mg IV: Participants who received risankizumab with inadequate response in Induction 1 randomized to receive risankizumab 1800mg administered by intravenous (IV) infusion in Induction 2.
  1 subject was dosed differently in period S1P1 (assigned to Pbo IV but dosed with Risa 600mg IV). This subject was classified into Risa 1800mg IV vs IV PbO based on the treatment received in S1P1.
- Substudy 1, Induction Period 2: Double-blind Risankizumab 180mg SC: Participants who received risankizumab with inadequate response in Induction 1 randomized to receive risankizumab 180mg administered by subcutaneous (SC) injection in Induction 2.
  1 participant assigned to Risankizumab 180mg SC was dosed with Risankizumab 360mg SC and is counted in that arm.
- Substudy 1, Induction Period 2: Double-blind Risankizumab 360mg SC: Participants who received risankizumab with inadequate response in Induction 1 randomized to receive risankizumab 360mg administered by subcutaneous (SC) injection in Induction 2.
  1 participant assigned to Risankizumab 180mg SC was dosed with Risankizumab 360mg SC and is counted in this arm.
- Substudy 2, Induction Period 1: Double-blind Placebo IV: Participants randomized to receive placebo for risankizumab administered by intravenous (IV) infusion.
  1 participant assigned to Placebo IV was dosed with Risankizumab 1200mg IV and is counted in that arm.
- Substudy 2, Induction Period 1: Double-blind Risankizumab 1200mg IV: Participants randomized to receive risankizumab 1200mg administered by intravenous (IV) infusion.
  1 participant assigned to Placebo IV was dosed with Risankizumab 1200mg IV and is counted in this arm.
Arm/Group | Substudy 1, Induction Period 1: Double-blind Placebo IV | Substudy 1, Induction Period 1: Double-blind Risankizumab 600mg IV | Substudy 1, Induction Period 1: Double-blind Risankizumab 1200mg IV | Substudy 1, Induction Period 1: Double-blind Risankizumab 1800mg IV | Substudy 1, Induction Period 1: Openlabel Risankizumab 1800mg IV | Substudy 1, Induction Period 2: Double-blind Risankizumab 1800mg IV Pbo | Substudy 1, Induction Period 2: Double-blind Risankizumab 1800mg IV | Substudy 1, Induction Period 2: Double-blind Risankizumab 180mg SC | Substudy 1, Induction Period 2: Double-blind Risankizumab 360mg SC | Substudy 2, Induction Period 1: Double-blind Placebo IV | Substudy 2, Induction Period 1: Double-blind Risankizumab 1200mg IV | Substudy 2, Induction Period 2: Double-blind Risankizumab 1200mg IV Pbo | Substudy 2, Induction Period 2: Double-blind Risankizumab 1200mg IV | Substudy 2, Induction Period 2: Double-blind Risankizumab 180mg SC | Substudy 2, Induction Period 2: Double-blind Risankizumab 360mg SC
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/62 | 0/61 | 0/58 | 0/341 | 0/36 | 0/37 | 0/71 | 0/71 | 0/324 | 1/653 | 0/174 | 0/68 | 0/71 | 0/71
Serious Adverse Events (participants affected / at risk) | 6/59 | 6/62 | 4/61 | 5/58 | 25/341 | 3/36 | 1/37 | 6/71 | 7/71 | 34/324 | 17/653 | 4/174 | 1/68 | 4/71 | 1/71
Other Adverse Events (participants affected / at risk) | 14/59 | 13/62 | 12/61 | 12/58 | 76/341 | 11/36 | 6/37 | 4/71 | 16/71 | 64/324 | 101/653 | 23/174 | 9/68 | 10/71 | 23/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Substudy 1, Induction Period 1: Double-blind Placebo IV (N=59) | Substudy 1, Induction Period 1: Double-blind Risankizumab 600mg IV (N=62) | Substudy 1, Induction Period 1: Double-blind Risankizumab 1200mg IV (N=61) | Substudy 1, Induction Period 1: Double-blind Risankizumab 1800mg IV (N=58) | Substudy 1, Induction Period 1: Openlabel Risankizumab 1800mg IV (N=341) | Substudy 1, Induction Period 2: Double-blind Risankizumab 1800mg IV Pbo (N=36) | Substudy 1, Induction Period 2: Double-blind Risankizumab 1800mg IV (N=37) | Substudy 1, Induction Period 2: Double-blind Risankizumab 180mg SC (N=71) | Substudy 1, Induction Period 2: Double-blind Risankizumab 360mg SC (N=71) | Substudy 2, Induction Period 1: Double-blind Placebo IV (N=324) | Substudy 2, Induction Period 1: Double-blind Risankizumab 1200mg IV (N=653) | Substudy 2, Induction Period 2: Double-blind Risankizumab 1200mg IV Pbo (N=174) | Substudy 2, Induction Period 2: Double-blind Risankizumab 1200mg IV (N=68) | Substudy 2, Induction Period 2: Double-blind Risankizumab 180mg SC (N=71) | Substudy 2, Induction Period 2: Double-blind Risankizumab 360mg SC (N=71)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD LOSS ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ARTERIOSCLEROSIS CORONARY ARTERY (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BASEDOW'S DISEASE (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CATARACT (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANAL FISTULA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANAL PROLAPSE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COLITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COLITIS ULCERATIVE (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 16 (17) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 16 (18) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
ENTERITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GASTRITIS EROSIVE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAEMATEMESIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HEPATIC CIRRHOSIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANAPHYLACTIC REACTION (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABSCESS LIMB (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANAL ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
APPENDICITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CLOSTRIDIUM DIFFICILE INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CYSTITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CYTOMEGALOVIRUS INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEVICE RELATED SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ENDOCARDITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ENTERITIS INFECTIOUS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ERYSIPELAS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LARGE INTESTINE INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LUNG ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PAROTID ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PHARYNGEAL ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA HAEMOPHILUS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA MYCOPLASMAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
POST PROCEDURAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RECTAL ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SALMONELLOSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FIBULA FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FOREARM FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
SKELETAL INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SKIN LACERATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAEMOGLOBIN DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COLORECTAL ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PITUITARY TUMOUR BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RENAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CEREBRAL MASS EFFECT (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIZZINESS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ADJUSTMENT DISORDER (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GENERALISED ANXIETY DISORDER (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MAJOR DEPRESSION (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SUICIDAL IDEATION (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CALCULUS URINARY (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NEPHROLITHIASIS (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RENAL COLIC (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RENAL FAILURE (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
UTERINE PROLAPSE (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ERYTHEMA NODOSUM (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PEMPHIGOID (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERTENSION (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PERIPHERAL ARTERY OCCLUSION (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Substudy 1, Induction Period 1: Double-blind Placebo IV (N=59) | Substudy 1, Induction Period 1: Double-blind Risankizumab 600mg IV (N=62) | Substudy 1, Induction Period 1: Double-blind Risankizumab 1200mg IV (N=61) | Substudy 1, Induction Period 1: Double-blind Risankizumab 1800mg IV (N=58) | Substudy 1, Induction Period 1: Openlabel Risankizumab 1800mg IV (N=341) | Substudy 1, Induction Period 2: Double-blind Risankizumab 1800mg IV Pbo (N=36) | Substudy 1, Induction Period 2: Double-blind Risankizumab 1800mg IV (N=37) | Substudy 1, Induction Period 2: Double-blind Risankizumab 180mg SC (N=71) | Substudy 1, Induction Period 2: Double-blind Risankizumab 360mg SC (N=71) | Substudy 2, Induction Period 1: Double-blind Placebo IV (N=324) | Substudy 2, Induction Period 1: Double-blind Risankizumab 1200mg IV (N=653) | Substudy 2, Induction Period 2: Double-blind Risankizumab 1200mg IV Pbo (N=174) | Substudy 2, Induction Period 2: Double-blind Risankizumab 1200mg IV (N=68) | Substudy 2, Induction Period 2: Double-blind Risankizumab 180mg SC (N=71) | Substudy 2, Induction Period 2: Double-blind Risankizumab 360mg SC (N=71)
ANAEMIA (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 2 (3) | 1 (1) | 12 (12) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 19 (21) | 21 (21) | 5 (5) | 1 (1) | 2 (2) | 6 (6)
COLITIS ULCERATIVE (Gastrointestinal disorders) | 5 (6) | 1 (1) | 3 (3) | 1 (1) | 12 (12) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 17 (17) | 10 (10) | 3 (3) | 1 (1) | 3 (3) | 0 (0)
HAEMORRHOIDS (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (6) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
BRONCHITIS (Infections and infestations) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 19 (19) | 30 (30) | 10 (10) | 4 (4) | 4 (4) | 6 (6)
NASOPHARYNGITIS (Infections and infestations) | 4 (5) | 5 (5) | 3 (5) | 5 (6) | 24 (26) | 2 (2) | 4 (5) | 1 (1) | 6 (6) | 8 (9) | 18 (18) | 3 (3) | 0 (0) | 1 (1) | 4 (4)
PHARYNGITIS (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SINUSITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 2 (3) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 3 (4) | 2 (2) | 3 (3) | 4 (5) | 22 (25) | 2 (2) | 0 (0) | 2 (2) | 5 (5) | 7 (8) | 19 (25) | 3 (3) | 2 (4) | 1 (1) | 6 (6)
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2022-12-16): https://cdn.clinicaltrials.gov/large-docs/48/NCT03398148/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-10): https://cdn.clinicaltrials.gov/large-docs/48/NCT03398148/SAP_001.pdf